# **Polichem**

Protocol No.: PM1541

A Multicenter, Randomized, Double-blind, Parallel-Group, Controlled Study, to Assess The Efficacy and Safety of P-3074 Cutaneous Spray Solution, In The Treatment of Male Pattern Baldness



# STATISTICAL ANALYSIS PLAN

Version: Final 1.0
Date of Issue: 22-January-2018

Author: PPD

PPD

Polichem S.A Via Senago 42 D Lugano-Pazzallo CH-6912 Switzerland

Date of Issue: 22-January-2018

## **APPROVALS**

The undersigned agree that all required reviews of this document are complete, and approve this Statistical Analysis Plan as final. Programming of the tables, figures and listings based upon the specifications within this document can proceed.

| Covance Approval: | PPD |
|------------------------------|------|
| <u> </u> | |
| Signature | Date |
| PPD / Principal Statistician | |
| Printed Name/Title | |
| Polichem Annrovals | |
| | PPD |
| Signature | Date |
| PPD | |
| Printed Name/Title PPD | PPD |
| Signature PP | Date |
| PPD | |
| Printed Name/Title | |


Date of Issue: 22-January-2018 Polichem Protocol No. PM-1541

# **REVIEWERS**

The following reviews of the SAP were conducted:

| Name and Title | Role | Version Last | Company/ |
|---|---|---|---|
| | | Reviewed | Organization |
| PPD | Peer Review Statistician | Internal draft 1.0 | PPD |
| PPD | Lead Programmer | Internal draft 1.0 | PPD |
| PPD | Medical Writer | Internal draft 1.0 | PPD |
| PPD | Project Physician | Internal draft 1.0 | PPD |
| PPD | Project Manager | Internal draft 1.0 | PPD |
| PPD | Project Manager | External draft | Polichem |
| | | 0.1 | |
| PPD | Lead Statistician | External draft | Polichem |
| | | 0.1 | |
| PPD | Lead Statistician | External Final | Almirall |
| | | 1.0 working | |
| PPD | Lead Statistician | External Final | Polichem |
| | | 0.1 Dated on 06- | |
| | | Dec-2017 | |

# **VERSION HISTORY**

| Version Number | Version Date | Summary and rational of change(s) |
|---|---|---|
| External Final 1.0 - working | 30-Jun-2017 | Final working version before signed off |
| External Final 1.0 | 5-Dec-2017 | Final version to sign off |
| External Final 1.0 | 22-Jan-2018 | <ol> <li>CCI summary by number of recommended sprays</li> <li>Include Skin irritation incidence rate</li> <li>Final version to sign off</li> </ol> |

<sup>&</sup>lt;Only final versions of the SAP need to be recorded here.>

# **TABLE OF CONTENTS**

| AF | PRO | VALS | 2 |
|---|---|---|---|
| RF | EVIE | WERS | 3 |
| VE | ERSIC | ON HISTORY | 3 |
| GI | LOSS | ARY OF ABBREVIATIONS | 6 |
| 1 | | URCE DOCUMENTS | |
| 2 | | OTOCOL DETAILS | |
| _ | 2.1 | Study Objectives | |
| | 2.2 | Study Endpoints | |
| | 2.2 | 2.2.1 Primary Endpoint | |
| | | 2.2.2 Secondary Endpoints | |
| | | 2.2.3 Exploratory Endpoints | |
| | 2.3 | Overall Study Design | |
| | 2.4 | Sample Size and Power | |
| 3 | EFF | TCACY AND SAFETY VARIABLES | 8 |
| | 3.1 | Primary Efficacy Variables | |
| | 3.2 | Secondary Efficacy Variables | |
| | 3.3 | Safety Variables | |
| C | | | |
| S | ANA | ALYSIS POPULATIONS | 10 |
| Γ | 5.1 | All Randomized Population | |
| | 5.2 | Safety Population | |
| | 5.3 | Intent to Treat (ITT) Population | |
| | 5.4 | Per Protocol Population (PPP) | |
| | | 5.4.1 Important Protocol Violation Leading to Exclusion from the PPP Analysis | 10 |
| | CC | | |
| 6 | DAT | TA HANDLING | 11 |
| | 6.1 | Time points and Visit Windows | 11 |
| | 6.2 | Handling of Drop-outs or Missing Data | 11 |
| 7 | STA | TISTICAL METHODS | 12 |
| | 7.1 | General Principles | |
| | 7.3 | 1 | |
| | 7.2 | Subject Disposition and Data Sets Analyzed | 12 |
| | 7.2<br>7.3 | Protocol Violations | |
| | | | 13 |

**Version: Final 1.0**Polichem Protocol No. PM-1541

| Date of Issue: | <b>22-January-2018</b> |
|----------------|------------------------|
|----------------|------------------------|

PPD

| | | 7.4.2 | Prior and Concomitant Medications | 13 |
|---|---|---|---|---|
| | 7.5 | Measu | urements of Treatment Compliance | 14 |
| | | 7.5.1 | Compliance via Diary | 14 |
| | | 7.5.2 | Compliance via Return of Plastic Bottles/Capsules | 15 |
| | 7.6 | Effica | cy | 16 |
| | | 7.6.1 | Primary Efficacy Analysis | 16 |
| | | 7.6.2 | Secondary Efficacy Analysis | 17 |
| | | 7.6.3 | Sensitivity Analysis | 18 |
| | | 7.6.4 | Subgroup Analysis | 18 |
| | | CCI | | |
| | | CCI | | |
| | 7.7 | Safety | <i>y</i> | 19 |
| | | 7.7.1 | Extent of Exposure | 19 |
| | | 7.7.2 | Adverse Events | 20 |
| | | 7.7.3 | Skin Irritation | 21 |
| | | 7.7.4 | Laboratory Evaluations | 22 |
| | | 7.7.5 | Vital Signs | 23 |
| | | 7.7.6 | Physical Examination | 23 |
| | | 7.7.7 | Self-administered Sexual Dysfunction Questionnaire (IIEF-2) | 23 |
| | <b>7.8</b> | Interi | m Analysis | 24 |
| 8 | CHA | ANGES | S IN PLANNED ANALYSES | 24 |
| 9 | REF | EREN | CES | 24 |
| 10 | APP | ENDIC | CES | 25 |
| AP | PEN | DIX I - | - SCHEDULE OF EVENTS | 25 |
| | | | - TABLE, FIGURE AND LISTING SHELLS | |

Date of Issue: 22-January-2018

# **GLOSSARY OF ABBREVIATIONS**

| Abbreviation | Term |
|--------------|----------------------------------------------|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BCA | Best Case Analysis |
| BLQL | Below the Lower Quantification Limit |
| CI | Confidence Interval |
| CCI | |
| eCRF | Electronic Case report form |
| IMP | Investigational Medicinal Product |
| ITT | Intention-to-treat |
| LOCF | Last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MHGQ | Male Hair Growth Questionnaire |
| NC | Not Calculated |
| O.D. | Once Daily |
| PD | Pharmacodynamics |
| PK | Pharmacokinetics |
| PT | Preferred Term |
| PPP | Per Protocol Population |
| PTAE | Pre-Treatment Adverse Event |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SI units | International System of units |
| SOC | System Organ Class |
| TAHC | Target Area Hair Count |
| TEAE | Treatment-Emergent Adverse Event |
| TESAE | Treatment-Emergent Serious Adverse Event |
| WCA | Worst Case Analysis |

Version: Final 1.0 Date of Issue: 22-January-2018
Polichem Protocol No. PM-1541

## 1 SOURCE DOCUMENTS

The Statistical Analysis Plan (SAP) was written based on the following documentation:

| Document | Date | Version |
|--------------------|-------------|-------------------|
| Protocol Amendment | 8-Mar-2017 | Final Version 4.0 |
| <e>CRF</e> | 21-Sep-2017 | Version 4.0 |

### 2 PROTOCOL DETAILS

## 2.1 Study Objectives

The primary objective of this pivotal Phase III study is to determine whether 24 weeks of a daily treatment with P-3074, increases hair count in men with male pattern baldness compared to the vehicle.

## 2.2 Study Endpoints

## 2.2.1 Primary Endpoint

• Hair growth assessed by Target Area Hair Count (TAHC) in the vertex at 24 weeks.

## 2.2.2 Secondary Endpoints

- Hair growth assessed by TAHC in the vertex at 12 Weeks;
- Target Area Hair Width (TAHW) in the vertex at Weeks 12 and 24;
- Patient assessment in Male Hair Growth Questionnaire (MHGQ) Score at Weeks 12 and 24;
- Investigator Assessment of Improvement from Baseline to Week 12 and from Baseline to Week 24, assessed for vertex;
- Blind Assessor Assessment of Improvement from Baseline to Week 12 and from Baseline to Week 24, assessed for vertex;
- Assessment of sexual function at every visit (Sexual Function Index, IIEF-2);

PPD

- Assessment of adverse events (AEs) throughout the study:
- Assessment of the local tolerability by means of severity scores for skin irritation;

For the purpose of assessment of changes in hair growth by investigators and blind assessor, screening visits (where global photos are taken) will act as Baseline.

## 2.2.3 Exploratory Endpoints



## 2.3 Overall Study Design

This is a Phase III, multicenter, randomized, double-blind, double-dummy, parallel-group study. The aim is to evaluate the efficacy and safety of P-3074 cutaneous topical solution versus an active comparator of

Version: Final 1.0 Polichem Protocol No. PM-1541

Date of Issue: 22-January-2018

oral Finasteride in the treatment of the male pattern baldness across three treatment arms, in the ratio of 2:2:1 (A:B:C).

Group A: P-3074 o.d. + placebo of oral Finasteride 1 mg o.d.

Group B: P-3074 Vehicle + placebo of oral Finasteride 1 mg o.d.

Or

Group C: Finasteride 1 mg o.d. + P-3074 Vehicle

The study consists of a screening visit (Visit 1), a randomization visit (Visit 2), a treatment phase of 24 weeks (assessed at 4 or 12 week intervals) and a 1-month follow up.

## 2.4 Sample Size and Power

Group sample sizes of 144 patients randomized to P-3074 and 144 patients randomized to placebo achieve 99% power to detect superiority using a one-sided, two-sample t-test with a significance level (alpha) of the test equal to 0.025. The margin of superiority, i.e. the distance above the reference (placebo) mean that is required to be considered superior, is set to a 41 hair count while the true difference between P-3074 and placebo is assumed to be an 82 hair count and is estimated assuming a mean change from baseline to 6 months in hair count equal to -14 and +68 in placebo and P-3074 respectively. The data are drawn from populations with standard deviations (SD) of 88 in P-3074 and 75 in placebo.

Approximately 72 patients will be randomized to the active comparator arm (oral Finasteride 1 mg). Group sample sizes of 144 patients randomized to P-3074 and 72 patients randomized to oral Finasteride achieve a power close to one to reject the null hypothesis of equal serum col inhibition assuming a mean serum [CIIII] inhibition equal to 45.6 and 26.2 in oral Finasteride and P-3074 respectively, with a SD for both groups of 19.0(2) and with a significance level (alpha) of 0.050 using a two-sided two-sample equal-variance t-test.

Assuming an attrition rate equal to 20%, the total number of patients should be no less than 450 patients randomized to P-3074, placebo and oral Finasteride in a 2:2:1 allocation ratio. All computations were performed using PASS 13 Software.

#### 3 EFFICACY AND SAFETY VARIABLES

## 3.1 Primary Efficacy Variables

Total hair count after 24 weeks of treatment

## 3.2 Secondary Efficacy Variables

- Total hair count after 12 weeks of treatment
- Hair width after 12 and 24 weeks of treatment
- Patient assessment in Male Hair Growth questionnaire (MHGQ) at Weeks 12 and 24:
  - o Bald spot getting smaller

Date of Issue: 22-January-2018

- o Appearance of your hair
- o Growth of hair
- o Effectiveness in slowing down hair loss
- o The hair line at the front of your head
- o The hair line at the top of your head
- Overall assessed by a patient
- Score of Investigator Assessment of Improvement from Baseline to Week 12 and from Baseline to Week 24, assessed for vertex
- Score of Blind Assessment of Improvement from Baseline to Week 12 and from Baseline to Week 24, assessed for vertex

## 3.3 Safety Variables

- Adverse events (AEs)
- Physical examination
- Vital signs
- Clinical laboratory tests
  - Hematology

Hemoglobin concentration, hematocrit, red blood cell count and white blood cell count with differential and platelet count

o Clinical Chemistry

Transaminases (Aspartate aminotransferase [AST], Alanine aminotransferase [ALT]), total serum bilirubin (direct and indirect), gamma glutamyl transferase, alkaline phosphatase, serum creatinine, blood urea nitrogen, uric acid, glucose, potassium, calcium, chloride, testosterone, protein and albumin

Urinalysis

Protein content, glucose content, hemoglobin content, white blood cell content in sediment, red blood cell content in sediment, crystals content in sediment, casts content in sediment

- Local Tolerability/skin irritation
- Assessment of potential Sexual Dysfunction (IIEF-2):
  - o Erectile function score
  - o Orgasmic function score
  - Sexual desire score
  - o Intercourse satisfaction score
  - Overall satisfaction score



Date of Issue: 22-January-2018

• CCI

## 5 ANALYSIS POPULATIONS

A patient will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A patient will be defined as <u>eligible</u> if he meets all the inclusion/exclusion criteria. Otherwise he will be defined as a screening failure.

A patient will be defined as <u>enrolled</u> in the study if he is included in the interventional phase of the study. Enrolment will be performed through randomized allocation to a treatment arm/treatments sequence.

## 5.1 All Randomized Population

All enrolled patients who are randomized to a treatment group.

## **5.2** Safety Population

All randomized patients who receive at least one application of the investigational drug.

## 5.3 Intent to Treat (ITT) Population

All patients who have measurements in regards to hair count both at baseline and on treatment.

## 5.4 Per Protocol Population (PPP)

All patients in the ITT population

- who did not take forbidden medications;
- who complete the entire study without any major protocol violations.

Analysis done on the PPP will be considered supportive.

## 5.4.1 Important Protocol Violation Leading to Exclusion from the PPP Analysis

A blinded data review meeting will be set up when 100% of patients with clean data before last patient last visit are available but before unblinding. The meeting will focus on defining the final PPP for PPP analysis. Detail of exclusion criteria will be documented in the blinding review meeting report.



Date of Issue: 22-January-2018



### DATA HANDLING

## 6.1 Time points and Visit Windows

Day 1 is defined as the day of first treatment dose. Relative days after Day 1 are calculated as (assessment date – Day 1 date) + 1. Relative days prior to Day 1 are calculated as (assessment date – Day 1 date). The day prior to Day 1 is Day -1.

All relevant safety data will be analyzed using nominal study visits as defined in the Study Schedule and electronic case report form (eCRF). A visit window of 28 days will be applied to all efficacy endpoints at visit 5 and 15 days at visit 6. A scheduled assessment/photo shooting with valid readings will be used if it is available. If there is no valid efficacy assessment/photo shooting at a scheduled visit, the analysis window below (Table 1) will be applied to re-allocate a post baseline unscheduled assessment/photo reshoot with valid readings to a scheduled assessment/photo shooting.

Table 1 – Analysis window definition

| Scheduled visit post baseline | Targeted study day | Analysis window in study days |
|---|---|---|
| Week 12 (Visit 5) | 84 | 81 to 112 |
| Week 24 (Visit 6) | 168 | 165 to 183 |

## 6.2 Handling of Drop-outs or Missing Data

Assuming missing data follows Missing Completely At Random (MCAR) or a Missing At Random (MAR) mechanism, a maximum likelihood analysis on available data should theoretically induce less bias compared to commonly used and naïve imputation method such as LOCF. So, the mixed linear models for the main analyses described in section 7.6.1 will represent a suitable choice in handling missing data and correcting for the bias potentially caused by drop-outs in this study.

To assess the sensitivity of the results due to the presence of missing values; three supplemental analyses will be performed on the primary endpoint analysis:

- Last Observation Carried Forward (LOCF)<sup>[1]</sup>: Missing outcomes will be replaced by the last non-missing, post-baseline value. For example, if a patient withdraw from the study before Visit 6 (Week 24) but has available hair count data at the early withdrawal visit, then the data from the early withdrawal visit will be carried forward to Visit 6 (Week 24).
- Best Case Analysis (BCA)<sup>[1]</sup>: Missing post-baseline outcomes will be replaced by the best outcome (maximum hair count) within the same treatment group at any post-baseline measurement (including follow-up visit) during the study period.
- Worst Case Analysis (WCA)<sup>[1]</sup>: Missing post-baseline outcomes will be replaced by the worst outcome (minimum hair count) within the same treatment group at any post-baseline measurement (including follow-up visit) during the study period.

Handling of missing/incomplete AE start/stop date will be documented in Section 7.7.2 Adverse Events. .

Date of Issue: 22-January-2018

#### 7 STATISTICAL METHODS

## 7.1 General Principles

All data processing, summarization and analyses will be performed using the Hosted SAS Environment Version 9.3 (or later) of the SAS<sup>®</sup> statistical software package.

Unless specified otherwise, data will be displayed using the following treatment group labels, in the order presented:

- P-3074 + P
- Vehicle + P
- Vehicle + FNS

Where "P-3074 + P" represents P-3074 o.d. + placebo of oral Finasteride 1 mg o.d, "Vehicle + P" represents P-3074 Vehicle + placebo of oral Finasteride 1 mg o.d., and "Vehicle + FNS" represents Finasteride 1 mg o.d. + P-3074 Vehicle.

All data collected will be presented in listings by treatment group, country, subject, and visit (where applicable), unless otherwise specified.

Data will be presented in summary tables by treatment group and visit (where applicable). The category "Missing" will be presented if the number missing is greater than zero for at least one treatment group.

Descriptive summary statistics for continuous variables will include the number of subjects (N), mean, standard deviation (SD), median, first (Q1) and third (Q3) quartiles, minimum (Min) and maximum (Max).

Descriptive summary statistics for categorical variables will include frequency counts and percentages [n (%)]. Unless stated otherwise in the table shells, the denominator for percentage calculations will be the number of subjects in the analysis population.

Dates will be displayed as DDMMMYYYY.

All significance tests will be two-sided and use a 5% significance level accompanied with 95% confidence interval.

## 7.2 Subject Disposition and Data Sets Analyzed

Subject disposition will be based on all enrolled subjects and will be listed and summarized by treatment group and overall, and will include the number and percentage of subjects:

- with inform consent;
- screened:
- randomized;
- included in each study population (All Randomized, ITT, Safety, PPP, Colonia).

The number and percentage of subjects who complete the study and who discontinue early (before follow up visit), including a breakdown of the primary reasons for discontinuation, will be presented for the All Randomized Population.

A summary of the reasons for screen failure as well as the number of subjects screened but not randomized will be produced. No other information for screen failures will be presented.


The number and percentage of subjects in each country and each site will be presented for the Randomized Population.

## 7.3 Protocol Violations

All protocol violations will be listed and summarized by treatment group for the Randomized Population.

All important protocol violations from the ITT population leading to exclusion from the PPP (see Section 5.4.1) will be listed and summarized by treatment group.

## 7.4 Demographics and Other Baseline Characteristics

Demographic and baseline characteristics will be listed and summarized by treatment group and overall for ITT and Safety populations. Descriptive statistics will be presented for the continuous variables of:

- age (years) [calculated as (year of informed consent signed year of birth) and reported as integer;
- weight (kg);
- height (cm);
- body mass index (kg/m<sup>2</sup>) [calculated as (weight/height<sup>2</sup>) where weight is in kg and height is in m];

The total counts and percentages of subjects will be presented for the categorical variables of:

- race;
- ethnicity;
- current alcohol use;
- current smoking/tobacco use;
- smoke >=10 cigarettes/day
- drink >5 cups coffee/tea/day

No formal tests of statistical significance will be performed on the demographic and baseline data.

Other baseline measurements, such as vital signs and laboratory data will be summarized by treatment group with the post-baseline measurements.

## 7.4.1 Medical History

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) [Version 19.0]. All medical history will be listed, and the number and percentage of subjects with any medical history and the frequency and percentage of a medical history episode will be summarized for All Randomized Population by system organ class (SOC) and preferred term (PT) for each treatment group and overall.

Vertex pattern hair loss according to Norwood/Hamilton scale will also be listed and the number and percentage of subjects in each type will be summarized for both ITT and Safety Populations.

## 7.4.2 Prior and Concomitant Medications

Medications received prior to or concomitantly with treatment will be coded by PPD using the WHODrug Dictionary [Version MAR16B2E].


Prior medications and concomitant medications are defined as follows:

Prior medications are those taken with a start and stop date prior to the first day of study treatment.

Concomitant medications are those with a start date on or after the first dose date of treatment, or those with a start date before the first dose date of treatment and a stop date on or after the first dose date of treatment or ongoing at the end of the study period.

If there are missing/partial medication start/end dates, The following rule will be used to determine whether the medication is a concomitant medication:

- If month/year of the start date is after the month/year of Day 1, the medication will be considered as concomitant medication:
- If month/year of the start date is equal or before the month/year of Day 1, and the end date is present, the end date will be used to determine whether the medication is prior or concomitant. If the end date is on or after Study Day 1, the medication will be considered as concomitant medication. Otherwise, if the medication stopped before Study Day 1, then the medication is a prior medication.

If month/year of the start date is equal to the month/year of Day 1, and the end date is a partial date, the medication will be considered as concomitant medication.

If a medication cannot be classified as "prior" or "concomitant" after applying imputation rules for missing/incomplete dates, it will be classified as concomitant.

Prior medications and concomitant medications will be listed together and summarized separately by treatment for the ITT and Safety Populations.

The number and percentage of subjects using each medication will be displayed together with the number and percentage of subjects using at least one medication within each therapeutic class (ATC-Level 2) and generic term.

## 7.5 Measurements of Treatment Compliance

Based on the protocol, patient compliance should be 80-120%, based on the number of days treated. The percentage of compliant subjects will be presented for the ITT and Safety Populations.

## 7.5.1 Compliance via Diary

The patients enrolled will be asked to keep a diary to record their drug compliance on a daily basis. Data will be summarized by treatment group using descriptive statistics. Boxplots will be produced for treatment arm and methods of compliance calculations.

## 7.5.1.1 Compliance via Tablet

Compliance in percentage based on number of days treated with tablets will be calculated as follows:

Number of tablets actually taken based on the diary ×100% Number of tablets expected to be taken

Where number of tablets expected to be taken is calculated as:

(date of treatment discontinuation/date of treatment completion – date of first dose + 1)  $\times 1$ 


## 7.5.1.2 Compliance via Spray

Compliance in percentage based on number of days treated on spreads will be calculated as follows:

Where number of spray expected shots is calculated as:

(date of treatment discontinuation/date of treatment completion – date of first dose + 1) × Number of spray shots recommended per day

Summary statistics on the compliance via spray will be based on the number of spray instructed at the randomization visit.

## 7.5.2 Compliance via Return of Plastic Bottles/Capsules

## 7.5.2.1 Compliance via Tablets Returned

Compliance in percentage is based on the number of tablets dispensed and the number of tablets returned. On the eCRF compliance will be calculated as follows:

$$\frac{\text{Number of tablets taken based on the eCRF}}{\text{Number of tablets expected to be taken}} \times 100\%$$

Where number of tablets taken based on eCRF is calculated as:

Sum of (number dispensed – number returned)

Where number of tablets expected taken is calculated as:

(date of discontinuation/date of treatment completion – date of first dose + 1)  $\times 1$ 

## 7.5.2.2 Compliance via Bottles Returned

Compliance in percentage based on weight of bottles dispensed and returned recorded from vendor data will be calculated as follows:

$$\frac{\text{Net weight of solution used}}{\text{Expected weight solution used}} \times 100\%$$

Where expected weight of solution used is calculated as:

(date of discontinuation/date of treatment completion – date of first dose + 1) × Number of spray shots recommended per day  $\times$  0.05 ml  $\times$  0.91 g/cm<sup>3</sup>


Summary statistics on the compliance via bottle returned will be based on the number of spray instructed at the randomization visit.

Note: Missing returned bottle(s) is considered as not used and cannot be included in the net weight of solution used for compliance calculation.

Unused kits will have net weight of solution used as 0.

The percentage of compliance will then be summarized in the following categories:

- <80%
- $\geq 80\%$  and  $\leq 120\%$
- >120%

## 7.6 Efficacy

All primary, secondary efficacy analyses as well as sensitivity analysis will be summarized and analyzed for the ITT and PPP.

#### **Primary Efficacy Analysis** 7.6.1

The primary efficacy variable, i.e. the change in the hair count from baseline, will be summarized by visit and by treatment group using descriptive statistics. The primary efficacy variable will then be analyzed using the SAS PROC MIXED procedure.

The null hypothesis is that there is no difference between P-3074 and placebo in the mean change from baseline for the hair count at Visit 6 (Week 24).

The alternative hypothesis will be that there is a difference between P-3074 and placebo in the mean change from baseline for the hair count at Visit 6 (Week 24).

The primary efficacy data will be fitted by a mixed linear model for repeated measures with treatment (P-3074 or placebo), center, visit and the treatment-by-visit interaction as fixed effects and baseline hair count as a covariate. The variance-covariance matrix of unstructured form will be used in order to model the correlation between the two repeated measurements (over the post-baseline visits). In the case of a convergence problem with the unstructured covariance matrix, the following structures with robust sandwich estimator for the standard error of the fixed effect estimates will be assessed in a sequential fashion: heterogeneous Toeplitz, heterogeneous first-order autoregressive, Toeplitz, and compound symmetry. Maximum likelihood estimates of the treatment mean difference will be computed at Visit 6 (Week 24) together with the associated two-sided 95% confidence interval (CI) that will be calculated by using the Newton-Raphson algorithm implemented in the SAS® Mixed Procedure. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant. The interaction between treatment and center will be assessed. A two-sided p-value less than or equal to 0.10 will be considered statistically significant for the test of interaction between treatment and center. If a statistically significant interaction is observed, efforts will be made to determine whether and how the interaction may affect the treatment comparisons.

The pooling centers strategy to be used for the above mentioned models will be the following: Those centers with less than 10 patients that were randomized within the same country will be grouped as one big site for analysis to ensure the convergence of the. If the combined group is still less than 10 patients, it will then be grouped to the site with minimum number of patients randomized within the same country. In

Date of Issue: 22-January-2018 Version: Final 1.0 Polichem Protocol No. PM-1541

case that the model does not converge and after replacing the variance-covariance matrix as described in the paragraph above, sites with less than 15 patients will be gathered following the same strategy described. If the model failed to converge, the center effect will be replaced by the country effect (in case of not converging, any country with less than 15 patients, that country would be gathered with the niebougrhood country).

Same approach will be applied to all secondary efficacy analysis and sensitivity analysis.

Below is an SAS syntax example for primary analysis and secondary analyses.

## proc mixed;

```
class trt usubjid visit center;
   model chg = trt base visit center visit*trt;
   repeated visit/ type = un subject = usubjid ;
   lsmeans visit*trt/diff e cl;
quit;
```

Note: chg is change from baseline

The main analysis will be based on observed cases using the above mixed model only on ITT population. Supportive analysis will be based on observed cases only on PPP population. Detail of sensitivity analyses are described in section 7.6.3.

## 7.6.2 Secondary Efficacy Analysis

## **Total hair count after 12 weeks of treatment:**

Data will be summarized by visit by treatment group using descriptive statistics. The maximum likelihood estimate of the treatment mean difference at Visit 5 (Week 12) together with the associated two-sided 95% CI and p-value will be obtained through the mixed linear model employed for the primary endpoint analysis (see above).

Data will also be displayed graphically. Both the unadjusted and adjusted mean change from baseline over time by treatment will be presented.

## Hair width after 12 and 24 weeks of treatment:

Data will be summarized by visit by treatment group using descriptive statistics. Adjusted and Unadjusted mean hair width over time will also be plotted. Data will be fitted by a mixed linear model for repeated measures with treatment group, center, visit and treatment-by-visit interaction as fixed effects, baseline hair width as covariate, and with an unstructured variance-covariance matrix to take into account correlations among repeated measures within patient. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant.

## Self-administered MHGQ as assessed by the patient at Weeks 12 and 24:

No summary score is calculated. Each question is scored and analyzed individually. Data will be summarized by visit by treatment group using descriptive statistics for each question. Each question will be fitted by a mixed linear model for repeated measures with treatment group, center,


visit and treatment-by-visit interaction as fixed effects, and with an unstructured variancecovariance matrix to take into account correlations among repeated measures within patients. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant

## Blind assessor assessment of patient hair growth/loss change from baseline:

Data will be fitted by a mixed linear model for repeated measures with treatment group, center, visit and treatment-by-visit interaction as fixed effects and with an unstructured variancecovariance matrix to take into account correlations among repeated measures within patients. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant.

## Change from baseline in Investigator Assessment at 12 and 24 weeks:

Data will be summarized by visit by treatment group using descriptive statistics, and both adjusted unadjusted mean score over time will be plotted. Data will be fitted by a mixed linear model for repeated measures with treatment group, center, visit and treatment-by-visit interaction as fixed effects and with an unstructured variance-covariance matrix to take into account correlations among repeated measures within patients. Results will be reported as maximum likelihood estimates of the treatment difference at Weeks 12 and 24 together with associated two-tailed 95% CI. A two-sided test with a p-value less than or equal to 0.05 will be considered statistically significant.

## 7.6.3 Sensitivity Analysis

Sensitivity analyses will be based on the ITT and PPP and performed on the change in the hair count in 3 different approaches on missing data imputation as described in Section 6.2.

For each of the three sensitivity analyses (LOCF, BCA and WCA), the change in the hair count from baseline to Visit 5 (Week 12) will be fitted by a linear model with treatment arm (P-3074 or placebo), center and baseline value as covariates (analysis of covariance).

## 7.6.4 Subgroup Analysis

No Subgroup analysis will be performed for this study.

| CCI |
|-----|

Date of Issue: 22-January-2018

Date of Issue. 22-January



## 7.7 The SAS syntax example can is shown in 7.6.5. Safety

## 7.7.1 Extent of Exposure

Duration of overall exposure will be defined in days as for both tablets and spray use:

(date of last dose/spray shot whichever comes later – date of first dose/spray shot whichever comes earlier) + 1 – off-drug (where both form of drugs were not used) days

If the date of first dose date is missing, then date of first dose dispensed will be used. If last dose date is missing, then last known date of study treatment taken/shot will be used.

Duration of overall exposure will be listed and summarized using descriptive statistics for each treatment group for the ITT and Safety Populations.

Duration of tablet exposure will be defined in days as:

(date of last dose – date of first dose) + 1 – off-drug (tablets were not used) days

Duration of spray exposure will be defined in days as:

(date of last spray – date of first spray) + 1 – off-drug (spray were not used) days

Version: Final 1.0 Date of Issue: 22-January-2018
Polichem Protocol No. PM-1541

## 7.7.2 Adverse Events

All AEs recorded on the eCRF will be coded using the MedDRA dictionary [Version 19.0] and classified as either pre-treatment AEs (PTAEs) or treatment – emergent AEs (TEAEs) as follows:

- PTAEs: all AEs occurring before the first dose of the investigational medicinal product (IMP)
- TEAEs: all AEs occurring or worsening on or after the first dose of the IMP

In case of missing/partial AE start/end dates. The following decision rule will be performed:

- If month/year of the onset date is after the month/year of Day 1, the AE will be considered as a TEAE.
- If month/year of the onset date is equal to the month/year of Day 1, and the end date is present, the end date will be used to determine when the AE resolved. If the end date is on or after Study Day 1, the AE will be considered as TEAE; otherwise, if the AE stopped before Study Day 1, then it will be categorized as PTAE.
- If the month/year of the onset date is equal to the month/year of Day 1, and the end date is a partial date, the AE will be considered as TEAE.

If after implementing the above conventions, the onset date of the AE cannot be placed before, on, or after Day 1, then the event will be considered as TEAE.

All AE data will be listed by treatment group where treatment-emergence status will be flagged in the listing. Corresponding listings of serious TEAEs (SAEs), TEAEs leading to discontinuation of treatment and TEAEs resulting in death will be produced.

No summary table will be provided for PTAEs.

Summary tables of TEAEs by treatment group and overall will be produced for the Safety Population.

The intensity of all AEs is recorded as mild, moderate, or severe. If intensity is missing for a TEAE, it will be considered severe in the summary tables.

The relationship between an AE and treatment is assessed as related, possibly related, unlikely to be related, or not related. A treatment-related AE is an AE considered by the investigator as related or possibly related to treatment or with unknown/missing relationship to treatment.

An overview table will summarize the number and percentage of subjects with at least one of the following TEAEs, where subjects with more than one TEAE in a particular category are counted only once in that category:

- any TEAE;
- any TEAE by intensity (mild, moderate, severe);
- any TEAE leading to discontinuation from the study;
- Treatment-related TEAEs;
- Treatment-related TEAEs leading to discontinuation from the study;
- Treatment-emergent SAEs (TESAE);
- Treatment-related TESAEs;
- TESAEs leading to death;

PPD CONFIDENTIAL


Polichem Protocol No. PM-1541

PDD

Date of Issue: 22-January-2018

PPD

- Treatment-related TESAEs leading to death;
- TESAEs leading to discontinuation from the study;
- Treatment-related TESAEs leading to discontinuation from the study;

The number and percentage of subjects reporting each AE and the frequency and percentage of each reported AE will be summarized by SOC and PT for the Safety Population. Tables will be sorted alphabetically by SOC. PTs will be sorted by descending overall total. The following summaries will be produced:

- TEAEs, by SOC and PT;
- TEAEs related to treatment, by SOC and PT;
- TEAEs by relationship to treatment, by SOC and PT;
- TEAEs by maximum intensity, by SOC and PT;
- TEAEs related to treatment by maximum intensity, by SOC and PT;
- TEAEs causing discontinuation from the study, by SOC and PT;
- TEAEs related to treatment causing discontinuation from the study, by SOC and PT;
- TESAEs, by SOC and PT;
- TESAEs related to treatment, by SOC and PT;
- TEAEs leading to death, by SOC and PT.

In the above summaries, subjects with more than one AE within a particular SOC are counted only once for that SOC. Similarly, subjects with more than one AE within a particular PT are counted only once for that PT. For summaries by maximum intensity, subjects with multiple AEs within a particular SOC or PT will be counted under the category of their most severe AE within that SOC or PT. AEs with missing intensity will be included (as severe) with AEs within a particular SOC or PT.

No statistical comparisons of AEs between treatment groups will be performed.

## 7.7.3 Skin Irritation

The number and percentage of subjects reporting severity score for skin irritation will be listed displayed by treatment at Week 4, Week 8, Week 12, Week 24, Week 28 and early termination visit for the Safety Population in a summary table.

Event incidence rate will also be reported by treatment group during the treatment period as well as during the study period. Anything other than "No evidence of irritation" under Dermal Response will be considered as an Dermal Responsed Skin Irritation event. Anything other than "No other eveffects" under Other Effects will be considered as an Other Effects of Skin Irritation event.

Treatment period is considered as the duration between the first date and the last date of the study treatment. Events observed during the study treatment period will be summarized as the event incidence rate during the study treatment period.

Version: Final 1.0 Date of Issue: 22-January-2018
Polichem Protocol No. PM-1541

Study period is considered as the duration between the first date of the study treatment and patient's last date of contact. Events observed during the study period will be summarized as the event incidence rate during the study period.

A person may have more than 1 skin irritation events and number of events will be used to calculate the event incidence rate. A person may have more than one skin irritation events where number of events are used to calculate the event incidence rate.

Event incidence rate is calculated as the number of events interest devided by total personal time in years.

## 7.7.4 Laboratory Evaluations

Data for the hematology, blood chemistry, and urinalysis analyses listed below received from central laboratory will be listed and summarized in shift table by treatment group. If data for any additional analyses are also received then these will be listed only.

| Hematology | Serum Chemistry | Urinalysis |
|------------|-------------------------------|-----------------------|
| Hematocrit | Alanine aminotranferase (ALT) | Macroscopic analysis: |
| | · | |

All laboratory data will be reported in SI units. Out-of-reference-range values will be flagged as high (H) or low (L) in the listings.


Shift tables (i.e., cross-tabulations of below the lower limit of the normal range, within the limits of the normal range and above the upper limit of the normal range at baseline versus scheduled visits) will be presented where the reference ranges are available by treatment group for the Safety Population for each laboratory test including urinalysis test parameters that are reported qualitatively (e.g. glucose, proteins and urobilinogen). In addition, shift tables on urinalysis test parameters that are reported qualitatively will be presented by treatment group for the ITT Population.

For each laboratory analyte, the baseline value will be defined as the last scheduled or unscheduled value collected prior to the first dose of treatment. Assessments carried out on the day of first treatment administration are considered to have taken place before the treatment administration, if the corresponding times have not been recorded. For post-baseline, only data from scheduled visits and final visit will be included in the shift tables.

## 7.7.5 Vital Signs

The following vital signs will be listed and summarized by treatment group and visit:

- systolic and diastolic blood pressure (mmHg);
- heart rate (bpm);
- weight (kg);
- body temperature (°C).

Vital signs data will be listed and changes from baseline in vital signs will be summarized by visit and final visit using standard descriptive statistics for the ITT and Safety Populations. Body temperature will be recorded in both Celsius and Fahrenheit on the eCRF. For the reporting purpose, body temperature will be reported in Celsius. The baseline value will be defined as the last scheduled or unscheduled value collected prior to the first dose of treatment. Assessments carried out on day of first treatment administration are considered to have taken place before the treatment administration, if the corresponding times have not been recorded. For post-baseline, only data from scheduled visits will be included in the summary tables.

## 7.7.6 Physical Examination

The number and percentage of patients with physical examination abnormalities will be listed and presented by treatment at screening, Week 24, Week 28 and early termination visits for the ITT and Safety Populations in summary tables.

## **Self-administered Sexual Dysfunction Questionnaire (IIEF-2)**

A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The table below shows the association between each domain and its corresponding questions.

| Associate Questions | Max Score |
|---------------------|-------------------------------------------------|
| 1, 2, 3, 4, 5, 15 | 30 |
| 9, 10 | 10 |
| 11, 12 | 10 |
| 6, 7, 8 | 15 |
| 13, 14 | 10 |
| | 1, 2, 3, 4, 5, 15<br>9, 10<br>11, 12<br>6, 7, 8 |


Data will be listed and summarized for the ITT for each domain by treatment at each visit.

Each domain will be analysed through a mixed linear model for repeated measures with treatment group, center and visit and treatment-by-visit interaction as fixed effects, and with an unstructured variancecovariance matrix.

## 7.8 Interim Analysis

No interim analysis is planned.

## **CHANGES IN PLANNED ANALYSES**

Not applicable

#### 9 **REFERENCES**

CPMP. Points to Consider on Missing Data. EMEA: London, 2001. Available at 1 http://www.ema.europa.eu/docs/en GB/document library/Scientific guideline/2009/09/WC500 003641.pdf

Polichem Protocol No. PM-1541

Date of Issue: 22-January-2018
PPD

# 10 APPENDICES

# **Appendix I - Schedule of Events**

| | Screening | | Treatment Phase | | | | Follow up Phase (End of Study) | Early<br>Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|
| Visit | Visit 1 | Random<br>Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | |
| | -Week 2 | Day 1± 5d | Week<br>4±3d | Week<br>8±3d | Week<br>12±3d | Week<br>24±3d | Week 28±3d | |
| Patient's Informed<br>Consent Form signature | X | | | | | | | |
| Demographic and habits information | X | | | | | | | |
| Physical examination§ | X | | | | | X | X | X |
| Medical history/current diseases | X | | | | | | | |
| Prior and concomitant medication | X | | | | | | | |
| Vital signs | X | | | | | X | X | X |
| Check all<br>Inclusion/exclusion<br>criteria | X | X | | | | | | |
| Enrolment | X | | | | | | | |
| Dispense patient's card | X | | | | | | | |
| Global Photograph | X | | | | X | X | | X |
| Investigator assessment | X* | | | | X | X | | X |
| Blind Assessor (entry eligibility) | X | | | | | | | |
| Blind Assessor (efficacy) | X* | | | | X | X | | X |
| Safety Laboratory examinations | X | | | X | | X | | X |
| Check record | | X | X | X | X | X | X | X |

Polichem Protocol No. PM-1541

Date of Issue: 22-January-2018
PPD

| concomitant medication | | | | | | | |
|---|---|---|---|---|---|---|---|
| CCI | | | | | | | |
| CCI | | | | | | | |
| Macrophotography (hair count) | X | | | X | X | | X |
| MHGQ Questionnaire | | | | X | X | | X |
| Sexual Dysfunction <b>Questionnaire (IIEF-2)</b> | | X | X | X | X | X | X |
| Randomization | X | | | | | | |
| Dispense study medication | X | | | X | | | |
| Collect / return study medication | | X <sup>#</sup> | X <sup>#</sup> | X | X | | X |
| Drug Application at site | | X | X | X | X | | |
| Drug Compliance | | | | X | X | | X |
| Dispense study diary to the patient | X | | | | | | |
| Check of patient's study diary | | X | X | X | X | X | X |
| Collect / return study diary | | | | | | X | X |
| Severity score for skin irritation | | X | X | X | X | X | X |
| Record AEs | X | X | X | X | X | X | X |

<sup>\*</sup> Assessment of hair growth will be performed by investigator and blinded assessor at visits 5 and 6/EOT using global photographs as baseline

CCI

<sup>§</sup> Height will be measured only at screening

**Version: Final 1.0** Polichem Protocol No. PM-1541

Date of Issue: 22-January-2018

# **Appendix II - Table, Figure and Listing Shells**

The table, figure and listing shells and corresponding Table of Contents will be created in separate file but can be appended here for the paper copy of the SAP.

# TABLES, FIGURES, AND LISTINGS SHELLS

A Multicenter, Randomized, Double-blind, Parallel-Group, Controlled Study, to Assess The Efficacy and Safety of P-3074 Cutaneous Spray, Solution, In The Treatment of Male Pattern Baldness

TFL Status: Final 1.0 TFL Date: 2018-01-22T13:53:00

Study Drug: P-3074

Sponsor Reference:

PPD

## 1. INTRODUCTION

The table, figure, and listing (TFL) shells presented in this document are mock-ups and may be subject to minor format modifications once the actual data are used. The data represented in this document are used for example purposes only and do not reflect the actual study data captured. The overall contents in any individual TFL shell will not change, although additional tables may be added if necessary, thus changing the table number scheme. Significant changes will be approved by the responsible PPD Clinical Pharmacology project team member and communicated to the Sponsor.

# 1.1 General Programming Specifications

All TFLs will follow the following rules:

Papersize will be A4, with the following margins in Inches:

```
Landscape
top 1 left 1
bottom 1 right 1
```

Every TFL will have a footnote containing program location, name, run date and run time (optional).

Every TFL will have a header containing client name, protocol number and the status of the output.

Dry run – Draft – Final Draft – Final (others as needed)

Dates will be presented in the format DDMMMYYYY

The presentation order of the statistics will be:

n, Mean, SD, median, minimum, maximum. The abbreviations Med, Min, Max may be used, if necessary.

Rules for significant digits in safety data tables are as follows: if the raw value has x decimal places, then the mean, the median and the Q1 and Q3 will have x+1 decimal places, the standard deviation will have x+2 decimal places. A maximum if 5 decimal places will be displayed if it is a derived value or the raw value has more than 5 decimal places.

N will be presented as whole numbers.

Percentages will always be displayed with 1 decimal place.

All TFLs will be delivered in .pdf format.

## 1.2 Derived Parameters

Individual derived parameters (e.g. CCI parameters) and appropriate summary statistics will be reported to three significant figures.

## 1.3 Tables Summarizing Categorical Data

Tables that summarize categorical data will be created per these specifications:

- 1. If the number of events is zero, data will be presented as "No event".
- 2. All categories of a parameter will be included and displayed. If the categories of a parameter are ordered, all categories between the maximum possible category and the minimum category will be included, even if n=0 for a given category. If the categories are not ordered, all categories will be included even if n=0 for a given category.
- 3. A "missing" category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

## 2. TABLE OF CONTENTS

| | Overall Preface Tables, Figures and Listings | 8 |
|---|---|---|
| Table 14.1.1 | Summary of Disposition of Patients Overall | |
| Table 14.1.2 | Disposition of Patients by Country and Trial Site Randomized Population | 10 |
| Table 14.1.3 | Summary of Protocol Violations Randomized Population | |
| Table 14.1.4.1 | Summary of Demography ITT Population | |
| Table 14.1.4.2 | Summary of Demography Safety Population | |
| Table 14.1.5.1 | Summary of Medical History ITT Population | |
| Table 14.1.5.2 | Summary of Medical History Safety Population | 15 |
| Table 14.1.6.1 | Summary of Prior Medications ITT Population | |
| Table 14.1.6.2 | Summary of Prior Medications Safety Population | 16 |
| Table 14.1.7.1 | Summary of Concomitant Medications ITT Population | 17 |
| Table 14.1.7.2 | Summary of Concomitant Medications Safety Population | 17 |
| Table 14.1.8.1 | Summary of Treatment Compliance ITT Population | |
| Table 14.1.8.2 | Summary of Treatment Compliance Safety Population | 21 |
| Table 14.1.9.1 | Summary of Treatment Exposure ITT Population | 22 |
| Table 14.1.9.2 | Summary of Treatment Exposure Safety Population | 22 |
| Table 14.2.1.1 | Summary of Total Hair Count by Visit ITT Population | |
| Table 14.2.1.2 | Analysis of Change in Total Hair Count from Baseline after 12 and 24 Weeks of Treatment ITT Population | 26 |
| Table 14.2.2.1 | Summary of Total Hair Count by Visit PP Population | |
| Table 14.2.2.2 | Analysis of Change in Total Hair Count from Baseline after 12 and 24 Weeks of Treatment PP Population | 27 |
| Table 14.2.3.1 | Summary of Hair Width by Visit ITT Population | 24 |
| Table 14.2.3.2 | Analysis of Change in Hair Width from Baseline after 12 and 24 Weeks of Treatment ITT Population | 27 |
| Table 14.2.4.1 | Summary of Hair Width by Visit PP Population | |
| Table 14.2.4.2 | Analysis of Change in Hair Width from Baseline after 12 and 24 Weeks of Treatment PP Population | 27 |
| Table 14.2.5.1 | Summary of Self-administered (MHGQ) Score by Visit ITT Population | 29 |
| Table 14.2.5.2.1 | Analysis of Self-administered (MHGQ) Score - Bald Spot Getting Smaller as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population | 27 |
| Table 14.2.5.2.2 | Analysis of Self-administered (MHGQ) Score - Appearance of Your Hair as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population | 27 |
| Table 14.2.5.2.3 | Analysis of Self-administered (MHGQ) Score - Growth of Hair as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population | 27 |
| Table 14.2.5.2.4 | Analysis of Self-administered (MHGQ) Score - Effectiveness in Slowing Down Hair Loss as assessed by the Patient after 12 and 24 Weeks of Treatment ITT | |
| | Population | 27 |
| Table 14.2.5.2.5 | Analysis of Self-administered (MHGQ) Score - The Hair Line at the Front of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment ITT | |
| | Population | |
| Table 14.2.5.2.6 | Analysis of Self-administered (MHGQ) Score - The Hair on Top of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population | |
| Table 14.2.5.3 | Summary of Self-administered (MHGQ) Score by Visit PP Population | |
| Table 14.2.5.4.1 | Analysis of Self-administered (MHGQ) Score - Bald Spot Getting Smaller as assessed by the Patient after 12 and 24 Weeks of Treatment PP Population | |
| Table 14.2.5.4.2 | Analysis of Self-administered (MHGQ) Score - Appearance of Your Hair as assessed by the Patient after 12 and 24 Weeks of Treatment PP Population | |
| Table 14.2.5.4.3 | Analysis of Self-administered (MHGQ) Score - Growth of Hair as assessed by the Patient after 12 and 24 Weeks of Treatment PP Population | 28 |
| Table 14.2.5.4.4 | Analysis of Self-administered (MHGQ) Score - Effectiveness in Slowing Down Hair Loss as assessed by the Patient after 12 and 24 Weeks of Treatment PP | |
| | Population | 28 |
| Table 14.2.5.4.5 | Analysis of Self-administered (MHGQ) Score - The Hair Line at the Front of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment PP | |
| | Population | |
| Table 14.2.5.4.6 | Analysis of Self-administered (MHGQ) Score - The Hair on Top of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment PP Population | |
| Table 14.2.6.1 | Summary of Patient Hair Growth/Loss Assessed by Blind Assessor by Visit ITT Population | 24 |

| Table 14.2.6.2 | Analysis of Change in Patient Hair Growth/Loss Assessed by Blind Assessor ITT Population | 28 |
|---|---|---|
| Table 14.2.7.1 | Summary of Patient Hair Growth/Loss Assessed by Blind Assessor by Visit PP Population | |
| Table 14.2.7.2 | Analysis of Change in Patient Hair Growth/Loss Assessed by Blind Assessor PP Population | 28 |
| Table 14.2.8.1 | Summary of Patient Hair Growth/Loss Assessed by Investigator by Visit ITT Population | 30 |
| Table 14.2.8.2 | Analysis of Change in Patient Hair Growth/Loss Assessed by Investigator ITT Population | 28 |
| Table 14.2.9.1 | Summary of Patient Hair Growth/Loss Assessed by Investigator by Visit PP Population | 30 |
| Table 14.2.9.2 | Analysis of Change in Patient Hair Growth/Loss Assessed by Investigator PP Population | 20 |
| Table 14.2.10.1 | Summary of Self-administered (IIEF-2) Score by Visit ITT Population | |
| | Analysis of Change in Self-administered (IEF-2) Erectile Function Score ITT Population | |
| Table 14.2.10.2.1 | | |
| Table 14.2.10.2.2 | Analysis of Change in Self-administered (IIEF-2) Orgasmic Function Score ITT Population | |
| Table 14.2.10.2.3 | Analysis of Change in Self-administered (IIEF-2) Sexual Desire Score ITT Population | 28 |
| Table 14.2.10.2.4 | Analysis of Change in Self-administered (IIEF-2) Intercourse Satisfaction Score ITT Population | 28 |
| Table 14.2.10.2.5 | Analysis of Change in Self-administered (IIEF-2) Overall Satisfaction Score ITT Population | 28 |
| Table 14.2.10.3 | Summary of Self-administered (IIEF-2) Score by Visit PP Population | |
| Table 14.2.10.4.1 | Analysis of Change in Self-administered (IIEF-2) Erectile Function Score PP Population | |
| Table 14.2.10.4.2 | Analysis of Change in Self-administered (IIEF-2) Orgasmic Function Score PP Population | 28 |
| Table 14.2.10.4.3 | Analysis of Change in Self-administered (IIEF-2) Sexual Desire Score PP Population | 28 |
| Table 14.2.10.4.4 | Analysis of Change in Self-administered (IIEF-2) Intercourse Satisfaction Score PP Population | 28 |
| Table 14.2.10.4.5 | Analysis of Change in Self-administered (IIEF-2) Overall Satisfaction Score PP Population | 28 |
| Table 14.2.11.1 | Summary of Total Hair Count at Baseline to Week 12 (LOCF) ITT Population | 32 |
| Table 14.2.11.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (LOCF) ITT Population | 33 |
| Table 14.2.12.1 | Summary of Total Hair Count at Baseline to Week 12 (LOCF) PP Population | 32 |
| Table 14.2.12.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (LOCF) PP Population | 33 |
| Table 14.2.13.1 | Summary of Total Hair Count at Baseline to Week 12 (BCA) ITT Population | |
| Table 14.2.13.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (BCA) ITT Population | |
| Table 14.2.14.1 | Summary of Total Hair Count at Baseline to Week 12 (BCA) PP Population | |
| Table 14.2.14.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (BCA) PP Population | |
| Table 14.2.15.1 | Summary of Total Hair Count at Baseline to Week 12 (WCA) ITT Population | |
| Table 14.2.15.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (WCA) ITT Population | 33 |
| Table 14.2.16.1 | Summary of Total Hair Count at Baseline to Week 12 (WCA) PP Population | 32 |
| Table 14.2.16.2 | Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (WCA) PP Population | 33 |
| CCI | | |
| T 11 142 1 1 | | |
| Table 14.3.1.1 | Overall Frequency of Patients with Adverse Events Safety Population | |
| Table 14.3.1.2 | Summary of Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term Safety Population | |
| Table 14.3.1.3 | Summary of Treatment-Related Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term Safety Population | |
| Table 14.3.1.4 | Summary of Treatment Emergent Adverse Events by Relationship to Study Treatment by MedDRA System Organ Class and Preferred Term Safety Population | |
| Table 14.3.1.5 | Summary of Treatment Emergent Adverse Events by Maximum Intensity System Organ Class and Preferred Term Safety Population | 42 |

| Table 14.3.1.6 | Summary of Treatment-Related Treatment Emergent Adverse Events by Maximum Intensity, System Organ Class and Preferred Term Safety Population | 43 |
|---|---|---|
| Table 14.3.1.7 | Summary of Treatment Emergent Adverse Events Causing Discontinuation from Study by MedDRA System Organ Class and Preferred Term Safety Population | 39 |
| Table 14.3.1.8 | Summary of Treatment-Related Treatment Emergent Adverse Events Causing Discontinuation from Study by MedDRA System Organ Class and Preferred Term Safety Population | 40 |
| Table 14.3.1.9 | Summary of Treatment-Related Treatment Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term Safety Population | 40 |
| Table 14.3.1.10 | Summary of Adverse Events Leading to Death by MedDRA System Organ Class and Preferred Term Safety Population | 40 |
| Table 14.3.1.11 | Summary of Severity Score for Skin Irritation Safety Population | 44 |
| Table 14.3.1.12 | Incidence Rate of Severity Score for Skin Irritation Safety Population | 45 |
| Table Listing 14.3.2 | Serious Treatment Emergent Adverse Events Safety Population | 46 |
| Table 14.3.4.1 | Shift Table of Hematology Test Results Safety Population | 47 |
| Table 14.3.4.2 | Shift Table of Serum Chemistry Test Results Safety Population | |
| Table 14.3.4.3.1.1 | Shift Table of Urinalysis Test Results ITT Population | |
| Table 14.3.4.3.1.2 | Shift Table of Urinalysis Test Results Safety Population | 52 |
| Table 14.3.4.3.2.1 | Shift Table of Urinalysis Test Results ITT Population | |
| Table 14.3.4.3.2.2 | Shift Table of Urinalysis Test Results Safety Population | 40 |
| Table 14.3.4.3.3.1 | Shift Table of Urinalysis Test Results ITT Population | |
| Table 14.3.4.3.3.2 | Shift Table of Urinalysis Test Results Safety Population | 53 |
| | Summary of Vital Signs ITT Population | |
| Table 14.3.5.1<br>Table 14.3.5.2 | | |
| | Summary of Vital Signs Safety Population | 34 |
| Table 14.3.6.1 | Summary of Physical Exam ITT Population | 33 |
| Table 14.3.6.2 | Summary of Physical Exam Safety Population | |
| Listing 16.2.1.1 | Patients Screened All Screened Patients | 56 |
| Listing 16.2.1.2 | Patients Disposition All Randomized Population | |
| Listing 16.2.1.3 | Patients Disposition All Randomized Population | 58 |
| Listing 16.2.1.4 | Patients Treatment Allocation All Randomized Population | 59 |
| Listing 16.2.1.5 | Protocol Violations All Randomized Population | 60 |
| Listing 16.2.2.1 | Inclusion Criteria All Screened Patients | 61 |
| Listing 16.2.2.2 | Exclusion Criteria All Screened Patients | |
| Listing 16.2.3 | Study Population All Screened Patients | |
| Listing 16.2.4.1 | Demographics All Randomized Population | |
| Listing 16.2.4.2 | Medical History All Randomized Population | 65 |
| Listing 16.2.4.3 | Prior and Concomitant Medication All Randomized Population | 66 |
| Listing 16.2.5.1 | Study Drug Administration (Tablet) All Randomized Population | |
| Listing 16.2.5.2 | Study Drug Administration (Spray) All Randomized Population | |
| Listing 16.2.5.3 | Study Treatment Compliance/Exposure All Randomized Population | |
| Listing 16.2.6.1 | Hair Assessment Results All Randomized Population | 70 |
| Listing 16.2.6.2 | MHGQ Questionnaire All Randomized Population | 71 |
| Listing 16.2.6.3 | Blind Assessor Assessment of Patient Hair Growth/Loss Change from Baseline All Randomized Population | |
| Listing 16.2.6.4 | Investigator's Assessment of Patient Hair Growth/Loss Change from Baseline All Randomized Population | 72 |
| CCI | | |
| Listing 16.2.7.1 | Adverse Events Safety Population | 74 |
| C | Treatment Emergent Adverse Events Leading to Discontinuation of Treatment Safety Population | |
| Listing 16.2.7.2 | | |
| Listing 16.2.7.3 | Death Safety Population | |
| Listing 16.2.7.4 | Severity Score for Skin Irritation Safety Population | |
| Listing 16.2.8.1 | Preface to Laboratory Findings Safety Population | |
| Listing 16.2.8.2 | Laboratory Findings - Hematology Safety Population | |
| Listing 16.2.8.3 | Laboratory Findings - Serum Chemistry Safety Population | 77 |

| Listing 16.2.8.4 | Laboratory Findings - Urinalysis Safety Population | 78 |
|---|---|---|
| Listing 16.2.8.5 | Vital Signs Safety Population | 79 |
| Listing 16.2.8.6 | Physical Examination Results Safety Population | 80 |
| Listing 16.2.8.7 | Self-administered Sexual Dysfunction Questionnaire Safety Population | 81 |
| Figure 14.1.6 | Study Treatment Compliance ITT Population | 82 |
| Figure 14.2.1.1 | Hair Count Unadjusted Mean Change From Baseline by Treatment Over Time ITT Population | 83 |
| Figure 14.2.1.2 | Hair Count Adjusted Mean Change From Baseline by Treatment Over Time ITT Population | 83 |
| Figure 14.2.2.1 | Hair Count Unadjusted Mean Change From Baseline by Treatment Over Time PP Population | 83 |
| Figure 14.2.2.2 | Hair Count Adjusted Mean Change From Baseline by Treatment Over Time PP Population | 83 |
| Figure 14.2.3.1 | Hair Width Unadjusted Mean Change From Baseline by Treatment Over Time ITT Population | |
| Figure 14.2.3.2 | Hair Width Adjusted Mean Change From Baseline by Treatment Over Time ITT Population | 83 |
| Figure 14.2.4.1 | Hair Width Unadjusted Mean Change From Baseline by Treatment Over Time PP Population | 84 |
| Figure 14.2.4.2 | Hair Width Adjusted Mean Change From Baseline by Treatment Over Time PP Population | 84 |
| Figure 14.2.8.1 | Unadjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time ITT Population | 85 |
| Figure 14.2.8.2 | Adjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time ITT Population | 85 |
| Figure 14.2.9.1 | Unadjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time PP Population | 85 |
| Figure 14.2.9.2 | Adjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time PP Population | |
| Figure 14.2.4.10.1 | Plasma Finasteride Concentration by Treatment Over Time Safety Population | 86 |

# Overall Preface Tables, Figures and Listings

- Patient Excluded from Safety Population
- \$ Patient Excluded from Intent-to-Treat Population (ITT)
- & Patient Excluded from Per-Protocol Population
- (R) Repeat Visit
- (W) Patient Withdrew
- (M) Patient Misrandomized
- NA Not Applicable
- NC Not Calculated
- ND Not Done
- NK Not Known
- NR Not Recorded

Program Name: Date Generated: Page x of y

Table 14.1.1 Summary of Disposition of Patients Overall

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| Patients with Informed Consent | | | | XXX |
| Patients Screened | | | | XXX |
| Patients Randomized | XXX | XXX | XXX | XXX |
| Safety Population | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| ITT Population | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Per Protocol Population | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| CCI | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Completed Study | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Primary Reason for Early Discontinuati | on: | | | |
| Adverse Event | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Death | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Lack of Efficacy | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Lost to Follow-Up | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Non-Compliance with Study Drug | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Physician Decision | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Protocol Deviation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Study Terminated by Sponsor | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Site Terminated by Sponsor | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Technical Problems | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Withdrawal by Patient | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

The denominator for percentages is the number of patients in the All Randomized Population for each treatment group. Programming Notes:

Obtain reasons for early discontinuation from CRF. Counts for screened patients will only be presented in the total column. Program Name:

Date Generated:

Page x of y
Table 14.1.2
Disposition of Patients by Country and Trial Site
Randomized Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| German | · | | | |
| Site 1 name | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Site 2 name | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Site 3 name | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Total | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Grouped sites: xxx, yyy, zzz | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Hungary | | | | |
| Site 1 name | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| Site 2 name | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Site 3 name | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Total | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |

Note: Sites with less than 8 patients who are randomized within the same country will be grouped as one big site for analysis to ensure model converging. If the combined group is still less than 8 patients, it will then be grouped to the site with minimum number of patients randomized in the neighboring country.

## Programming Notes:

Only include "Grouped site" if number of patient in each individual site is less than 8 and grouping is required for modelling. Program Name:

Page x of y

Table 14.1.3
Summary of Protocol Violations
Randomized Population

| Protocol Violation | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| Patients with at Least 1 Major Protocol Violation | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Major Protocol Violation 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| etc | | | | |

The violations and deviations were identified prior to data unblinding.

Program Name: Date Generated:

Table 14.1.4.1
Summary of Demography
ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| Age (Years) [a] | | | | |
| n | XXX | xxx | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | xx.x | XX.XX |
| Q1, Q3 | XXX, XXX | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | xx.x | xx.xx |
| Max | xx.x | XX.X | XX.X | XX.XX |
| Height (cm) | | | | |
| n | XXX | xxx | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | xx.x | xx.xx |
| Q1, Q3 | XXX, XXX | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | XX.X | xx.x | XX.XX |
| Max | xx.x | XX.X | XX.X | XX.XX |
| Weight (kg) | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.XX |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X | XX.XX |
| Max | XX.X | XX.X | XX.X | XX.XX |

Note: Denominators for percentages are based on the number of patients with non-missing data in each treatment group for the relevant variable.
[a] Age is calculated as calendar years from birth to informed consent

Program Name: Date Generated: Page x of y

<sup>[</sup>b] Body Mass Index

Table 14.1.4.1 Summary of Demography ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = XXX) | (N = xxx) | (N = xxx) | (N = XXX) |
| BMI (kg/m2) [b] | | | | |
| n | xxx | xxx | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.xx |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | xx.x | XX.X | XX.XX |
| Max | XX.X | XX.X | XX.X | XX.XX |
| ace, n (%) | | | | |
| n | xxx | XXX | XXX | xxx |
| Asian | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Black/African American | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Caucasian/White | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Native Hawaiian/Pacific Islander | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| American Indian/Alaska Native | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Other | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Ethnicity, n (%) | | | | |
| n | xxx | xxx | xxx | xxx |
| Hispanic or Latino | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| Not Hispanic or Latino | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| Not Provided or Unknown | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

Note: Denominators for percentages are based on the number of patients with non-missing data in each treatment group for the relevant variable. [a] Age is calculated as calendar years from birth to informed consent

Program Name: Date Generated: Page x of y

<sup>[</sup>b] Body Mass Index

Table 14.1.4.1 Summary of Demography ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| urrent Alcohol Use, n(%) | | | | |
| n | XXX | xxx | XXX | XXX |
| None | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Less Than or Equal to 2 Drinks<br>Per Day | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| More Than 2 Drinks Per Day | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| rrent Smoke/Tobacco Use, n (%) | | | | |
| n | XXX | XXX | XXX | XXX |
| Never Smoked/Never Used Tobacco<br>Products | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Currently Smokes/Uses Tobacco<br>Products | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Formally Smoked/Used Tobacco<br>Product | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| oke >=10 Cigarettes/Day, n (%) | | | | |
| n | xxx | XXX | XXX | xxx |
| Yes | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| No | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| ink > 5 Cup Coffee/Tea/Day, n (%) | | | | |
| n | XXX | XXX | XXX | XXX |
| Yes | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| No | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

Note: Denominators for percentages are based on the number of patients with non-missing data in each treatment group for the relevant variable.

[a] Age is calculated as calendar years from birth to informed consent

Program Name: Date Generated:

Repeat for the following displays:

Table 14.1.4.2 Summary of Demography Safety Population

<sup>[</sup>b] Body Mass Index

Table 14.1.5.1
Summary of Medical History
ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) |
| Vertex Pattern Hair Loss | According to Norwood/Hamilt | con Scale | | |
| Type III Vertex | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Type IV | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Type V | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Other | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Patients with Any Curren | t Medical History? | | | |
| No | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Yes | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Medical History | | | | |
| System Organ Class 1 | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 1 | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 2 | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 3 | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 4 | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| System Organ Class 1 | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| | 1 11/2 1 11 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| : | xxx(xx.x%)/xxx(xx.x%) | XXX (XX.X6) / XXX (XX.X6) | AAA (AA • A o ) / AAA (AA • A o ) | AAA (AA • A o ) / AAA (AA • A o ) |

n = number of patients in each category; The percentage is calculated as 100 x (n/N)

Note: MedDRA Version MAR16B2E used for coding.

Program Name: Date Generated:

Repeat for the following displays:

Table 14.1.5.2 Summary of Medical History Safety Population

e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

Note: This table contains counts of patients. If a patient had more than one medical history within a preferred term, the patient is counted only once within a preferred term. If a patient had more than one medical history within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Table 14.1.6.1
Summary of Prior Medications
ITT Population

| WHO ATC Level 2 (Therapeutic Class) | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| Generic Term ([a]) | (N = xxx) | (N = xxx) | (N = xxx) | (N = XXX) |
| Patients with Any Prior Medication? | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| ATC Level 2 Term 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Generic Medication 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 3 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 4 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| ATC Level 2 Term 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 3 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 4 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

The denominator for percentages is the number of patients in the ITT Population for each treatment group.

Note: Prior medications are defined as medications taken with a start and stop date prior to the first day of study treatment.

Note: A patient may have taken more than one medication. Therefore, the sum of medication counts and percentages may not equal the total counts.

If a patient had more than one medication in a category, the patient is counted once in that category.

[a] WHO Drug Dictionary (Version MAR16B2E) was used for coding.

Program Name: Date Generated:

Repeat for the following displays:

Table 14.1.6.2 Summary of Prior Medications Safety Population

Add:

Footnote: The denominator for percentages is the number of patients in the Safety Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients in the ITT Population for each treatment group.

Table 14.1.7.1
Summary of Concomitant Medications
ITT Population

| WHO ATC Level 2 (Therapeutic Class) Generic Term ([a]) | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| Patients with Any Concomitant Medication? | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| ATC Level 2 Term 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 1 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 3 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 4 | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| ATC Level 2 Term 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 1 | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Generic Medication 2 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Generic Medication 3 | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Generic Medication 4 | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

The denominator for percentages is the number of patients in the ITT Population for each treatment group.

Note: Concomitant medications are defined as medications taken with a start date on or after the first dose date of treatment, or those with a start date before the first dose date of treatment and a stop date on or after the first dose date of treatment or ongoing at the end of the study period.

Note: A patient may have taken more than one medication. Therefore, the sum of medication counts and percentages may not equal the total counts.

If a patient had more than one medication in a category, the patient is counted once in that category.

[a] WHO Drug Dictionary (Version MAR16B2E) was used for coding.

Program Name: Date Generated:

Repeat for the following displays:

Table 14.1.7.2 Summary of Concomitant Medications Safety Population

Add:

Footnote: The denominator for percentages is the number of patients in the Safety Population for each treatment group.

## Delete:

Footnote: The denominator for percentages is the number of patients in the ITT Population for each treatment group.

Table 14.1.8.1
Summary of Treatment Compliance
ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = XXX) | (N = xxx) | (N = xxx) | (N = xxx) |
| ompliance Via Diary(%) | | | | |
| Tablets Count | | | | |
| n | XXX | xxx | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | xx.x | xx.xx |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | xx.x | xx.x | XX.XX |
| Max | XX.X | XX.X | XX.X | xx.xx |
| <80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| 80% to 120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| >120% | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Actual spray count for those prescribed | | | | |
| with 1 Spray | | | | |
| n | XXX | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X | XX.XX |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | XX.X | XX.X | XX.XX |
| Max | XX.X | XX.X | XX.X | XX.XX |

<repeat for 2 sprays, 3 sprays and 4
sprays>

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group. Compliant is defined as percentage compliance between 80.0% and 120.0%, inclusive.

Program Name:

Date Generated:

Page x of y

Table 14.1.8.1
Summary of Treatment Compliance
ITT Population

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| anon Compliano | · | | | . , , |
| oray Compliance<br>Ompliance among with those wit | ch 1 Spray prescribed | | | |
| - | | | | |
| < 80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| 80% to 120% | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| >120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| repeat for 2 sprays, 3 sprays | and 4 sprays> | | | |
| ompliance among with those wit | th 1-4 Spray prescribed | | | |
| <80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| 80% to 120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| >120% | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group. Compliant is defined as percentage compliance between 80.0% and 120.0%, inclusive.

Program Name: Date Generated: Page x of y

Table 14.1.8.1
Summary of Treatment Compliance
ITT Population

| | P-3074 + P $(N = xxx)$ | <pre>Vehicle + P (N = xxx)</pre> | Vehicle + FNS<br>(N = xxx) | Overall Total $(N = xxx)$ |
|---|---|---|---|---|
| ompliance Via Drug Accountability(%) | | | | |
| Tablets Count | | | | |
| n | XXX | xxx | XXX | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | XX.X | xx.xx |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | xx.x | xx.x | xx.x | XX.XX |
| Max | XX.X | XX.X | XX.X | XX.XX |
| <80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| 80% to 120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| >120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Bottle Weight-1 Spray | | | | |
| n | xxx | xxx | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | XX.X | XX.XX |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | xx.x | xx.x | XX.X | XX.XX |
| Max | XX.X | xx.x | xx.x | xx.xx |

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group. Compliant is defined as percentage compliance between 80.0% and 120.0%, inclusive.

Program Name:

Date Generated:

Page x of y

Table 14.1.8.1
Summary of Treatment Compliance
ITT Population

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| Compliance Bottle Weight-1 Spray | | | | |
| <80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| 80% to 120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| >120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Repeat for Bottle Weight-2 Spray, 3 s | prays and 4 sprays> | | | |
| Compliance Bottle Weight-1-4 Spray | | | | |
| <80% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| 80% to 120% | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| >120% | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group. Compliant is defined as percentage compliance between 80.0% and 120.0%, inclusive.

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.1.8.2 Summary of Treatment Compliance Safety Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the Safety Population for each treatment group.

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.1.9.1
Summary of Treatment Exposure
ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| Duration (days) | | | |
| n | xxx | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | xx.x |
| Max | XX.X | XX.X | XX.X |
| Duration of tablets exposure(days) | | | |
| n | XXX | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |
| Duration of spray exposure(days) | | | |
| n | XXX | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |

Duration of overall exposure is calculated as (date of last dose/spray shot whichever comes later - date of first dose/spray shot whichever comes earlier) + 1 - off-drug (where both form of drugs were not used) days.

Duration of table exposure is calculated as (date of last dose - date of first dose) + 1 - off-drug (tablets were not used) days. Duration of spray exposure is calculated as (date of last spray - date of first spray) + 1 - off-drug (spray were not used) days. Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.1.9.2 Summary of Treatment Exposure Safety Population

Footnote: The denominator for percentages is the number of patients with non missing data in the Safety Population for each treatment group.

Duration of overall exposure is calculated as (date of last dose/spray shot whichever comes later - date of first dose/spray shot whichever comes earlier) + 1 - off-drug (where both form of drugs were not used) days.

Delete:

Footnote: Duration of overall exposure is calculated as (date of last dose/spray shot whichever comes later - date of first dose/spray shot whichever comes earlier) + 1 - off-drug (where both form of drugs were not used) days.

Table 14.2.1.1
Summary of Total Hair Count by Visit ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS |
|----------------------|---------------|---------------|----------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| aseline | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |
| Visit> | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XXX, XXX | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |
| Change from Baseline | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | xx.x | XX.X |

[Repeat for all scheduled visits]

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.2.1 Summary of Total Hair Count by Visit PP Population

Table 14.2.3.1 Summary of Hair Width by Visit ITT Population

Table 14.2.4.1 Summary of Hair Width by Visit PP Population

Table 14.2.6.1 Summary of Patient Hair Growth/Loss Assessed by Blind Assessor by Visit ITT Population

Table 14.2.7.1 Summary of Patient Hair Growth/Loss Assessed by Blind Assessor by Visit PP Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| Number of patients | XXX | XXX | XXX |
| Baseline Unadjusted Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| 12 Weeks Visit | | | |
| Unadjusted Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Unadjusted Mean Change from Baseline(SE) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Adjusted Mean Change from Baseline(SE)[a] | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Versus P-3074 + P | | | |
| LS Mean Difference (SE) [a] | | x.xx (x.xxx) | |
| 95% Confidence Interval [a] | | (x.xx, x.xx) | |
| p-value [a] | | X.XXX | |

<sup>[</sup>a] The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects and baseline hair count as a covariate with an unstructured covariance structure. Change from Baseline by Visit is the reported result.

Program Name:

Date Generated:

Page x of y

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) |
|---|---|---|---|
| 24 Weeks Visit | | | |
| Unadjusted Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Unadjusted Mean Change from Baseline(SE) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Adjusted Mean Change from Baseline(SE)[a] | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Versus P-3074 + P | | | |
| LS Mean Difference (SE) [a] | | x.xx (x.xxx) | |
| 95% Confidence Interval [a] | | (x.xx, x.xx) | |
| p-value [a] | | X.XXX | |

[a] The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects and baseline hair count as a covariate with an unstructured covariance structure. Change from Baseline by Visit is the reported result.

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.2.2.2 Analysis of Change in Total Hair Count from Baseline after 12 and 24 Weeks of Treatment PP Population

Table 14.2.3.2 Analysis of Change in Hair Width from Baseline after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.4.2 Analysis of Change in Hair Width from Baseline after 12 and 24 Weeks of Treatment PP Population

Table 14.2.5.2.1 Analysis of Self-administered (MHGQ) Score - Bald Spot Getting Smaller as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.5.2.2 Analysis of Self-administered (MHGQ) Score - Appearance of Your Hair as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.5.2.3 Analysis of Self-administered (MHGQ) Score - Growth of Hair as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.5.2.4 Analysis of Self-administered (MHGQ) Score - Effectiveness in Slowing Down Hair Loss as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.5.2.5 Analysis of Self-administered (MHGQ) Score - The Hair Line at the Front of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

Table 14.2.5.2.6 Analysis of Self-administered (MHGQ) Score - The Hair on Top of Your Head as assessed by the Patient after 12 and 24 Weeks of Treatment ITT Population

| Table 14.2.5.4.1 Treatment PP Populati | Analysis of Self-administered (MHGQ) Score - Bald Spot Getting Smaller as assessed by the Patient after 12 and 24 Weeks of on |
|---|---|
| Table 14.2.5.4.2 Treatment PP Populati | Analysis of Self-administered (MHGQ) Score - Appearance of Your Hair as assessed by the Patient after 12 and 24 Weeks of on |
| Table 14.2.5.4.3 PP Population | Analysis of Self-administered (MHGQ) Score - Growth of Hair as assessed by the Patient after 12 and 24 Weeks of Treatment |
| Table 14.2.5.4.4 and 24 Weeks of Treat | Analysis of Self-administered (MHGQ) Score - Effectiveness in Slowing Down Hair Loss as assessed by the Patient after 12 ment PP Population |
| Table 14.2.5.4.5<br>and 24 Weeks of Treat | Analysis of Self-administered (MHGQ) Score - The Hair Line at the Front of Your Head as assessed by the Patient after 12 ment PP Population |
| Table 14.2.5.4.6 of Treatment PP Popul | Analysis of Self-administered (MHGQ) Score - The Hair on Top of Your Head as assessed by the Patient after 12 and 24 Weeks ation |
| Table 14.2.6.2 Analys | is of Change in Patient Hair Growth/Loss Assessed by Blind Assessor ITT Population |
| Table 14.2.7.2 Analys | is of Change in Patient Hair Growth/Loss Assessed by Blind Assessor PP Population |
| Table 14.2.8.2 Analys | is of Change in Patient Hair Growth/Loss Assessed by Investigator ITT Population |
| Table 14.2.9.2 Analys | is of Change in Patient Hair Growth/Loss Assessed by Investigator PP Population |
| Table 14.2.10.2.1 | Analysis of Change in Self-administered (IIEF-2) Erectile Function Score ITT Population |
| Table 14.2.10.2.2 | Analysis of Change in Self-administered (IIEF-2) Orgasmic Function Score ITT Population |
| Table 14.2.10.2.3 | Analysis of Change in Self-administered (IIEF-2) Sexual Desire Score ITT Population |
| Table 14.2.10.2.4 | Analysis of Change in Self-administered (IIEF-2) Intercourse Satisfaction Score ITT Population |
| Table 14.2.10.2.5 | Analysis of Change in Self-administered (IIEF-2) Overall Satisfaction Score ITT Population |
| Table 14.2.10.4.1 | Analysis of Change in Self-administered (IIEF-2) Erectile Function Score PP Population |
| Table 14.2.10.4.2 | Analysis of Change in Self-administered (IIEF-2) Orgasmic Function Score PP Population |
| Table 14.2.10.4.3 | Analysis of Change in Self-administered (IIEF-2) Sexual Desire Score PP Population |
| Table 14.2.10.4.4 | Analysis of Change in Self-administered (IIEF-2) Intercourse Satisfaction Score PP Population |
| Table 14.2.10.4.5 | Analysis of Change in Self-administered (IIEF-2) Overall Satisfaction Score PP Population |

Table 14.2.5.1
Summary of Self-administered (MHGQ) Score by Visit
ITT Population

| Bald Spot Getting Smaller as Assessed by the Patient | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) |
|---|---|---|---|
| <visit></visit> | | | |
| Since the start of the study, I can see my bald spot getting smaller. | | | |
| Strongly agree (1) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Agree (2) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| No Opinion either way (3) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Disagree (4) | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Strongly disagree (5) | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Score | | | |
| n | XXX | xxx | xxx |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |

[Repeat for all scheduled visits]

Note: A higher score indicates a worse outcome.

Programming Notes:

Include Bald Spot Getting Smaller as Assessed by the Patient, Appearance of My Hair as Assessed by the Patient, Growth of Hair as Assessed by the Patient, Effectiveness in Slowing Down Hair Loss as Assessed by the Patient, The Hair Line at the Front of Your Head as Assessed by the Patient, The Hair on Top of Your Head as Assessed by the Patient, and Overall as Assessed by the Patient. Start with a new page with a new a new question from the questionnaire to be summarized.

Please note, each question has it own number of options to be choosen and wording to be displayed. Please cross check with the original questionnaire with correct wording and number selection options.

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.2.5.3 Summary of Self-administered (MHGQ) Score by Visit PP Population Delete:

Delete:

Note to Programmer: Please note, each question has it own number of options to be choosen and wording to be displayed. Please cross check with the original questionnaire with correct wording and number selection options.

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) |
|---|---|---|---|
| <visit></visit> | | | |
| ssessment of hair growth | | | |
| Greatly decreased (- | -3) xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Moderately decreased | d (-2) xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Slightly decreased | (-1) xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| No change (0) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Slightly increased | (1) xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Moderately increased | d (2) xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Greatly increased (3 | 3) xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Score | | | |
| n | xxx | XXX | XXX |
| Mean (SD) | xx.x ( xx.x | x) xx.x ( xx.xx | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XXX, XXX | xxx, xxx | xxx, xxx |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | xx.x |

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.9.1 Summary of Patient Hair Growth/Loss Assessed by Investigator by Visit PP Population

Table 14.2.10.1
Summary of Self-administered (IIEF-2) Score by Visit
ITT Population

| IIEF-2 Erectile Function Score | P-3074 + P | Vehicle + P | Vehicle + FNS |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| leek 4 | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | xx.x | xx.x | XX.X |
| Max | XX.X | XX.X | xx.x |
| Week 8 | | | |
| n | xxx | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | XX.X | XX.X | XX.X |
| Max | XX.X | XX.X | XX.X |

[Repeat for all IIEF-2 scheduled visits]

## Programming Notes:

Include IIEF-2 Erectile Function Score, IIEF-2 Orgasmic Function Score, IIEF-2 Sexual Desire Score, IIEF-2 Intercourse Satisfaction score, and IIEF-2 Overall Satisfaction Score. Start with a new page with a new function domain from the IIEF-2 questionnaire to be summarized.

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.2.10.3 Summary of Self-administered (IIEF-2) Score by Visit PP Population

Note to Programmer: Include IIEF-2 Erectile Function Score, IIEF-2 Orgasmic Function Score, IIEF-2 Sexual Desire Score, IIEF-2 Intercourse Satiscation score, and IIEF-2 Overall Satisfaction Score. Start with a new page with a new function domain from the IIEF-2 questionnaire to be summarized.

Delete:

Note to Programmer: Include IIEF-2 Erectile Function Score, IIEF-2 Orgasmic Function Score, IIEF-2 Sexual Desire Score, IIEF-2 Intercourse Satisfaction score, and IIEF-2 Overall Satisfaction Score. Start with a new page with a new function domain from the IIEF-2 questionnaire to be summarized.

| | | | 1 | | |
|---|---|---|---|---|---|
| | | P-3074 + P | Vehicle + P | Vehicle + FNS | · |
| | | (N = xxx) | (N = xxx) | (N = xxx) | |
| Baseline | | | | | |
| n | | XXX | XXX | XXX | |
| Mean (SD) | | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | |
| Median | | XX.X | XX.X | XX.X | |
| Q1, Q3 | | xxx, xxx | xxx, xxx | xxx, xxx | |
| Min | | XX.X | XX.X | XX.X | |
| Max | | XX.X | XX.X | XX.X | |
| Week 12 | | | | | |
| n | | xxx | XXX | XXX | |
| Mean (SD) | | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | |
| Median | | XX.X | XX.X | XX.X | |
| Q1, Q3 | | xxx, xxx | xxx, xxx | xxx, xxx | |
| Min | | XX.X | XX.X | XX.X | |
| Max | | XX.X | XX.X | XX.X | |
| Change from Baseli | ine | | | | |
| n | | XXX | XXX | XXX | |
| Mean (SD) | | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) | |
| Median | | xx.x | XX.X | XX.X | |
| Q1, Q3 | | xxx, xxx | xxx, xxx | xxx, xxx | |
| Min | | XX.X | xx.x | XX.X | |
| Max | | XX.X | XX.X | XX.X | |
| Program Name: | | Date Generat | ed: | | Page x of y |
| Repeat for the follo | owing displays: | | | | - |
| Table 14.2.12.1 | Summary of Total Ha | ir Count at Basel: | ine to Week 12 (LOCF | ) PP Population | |
| Table 14.2.13.1 | Summary of Total Ha | ir Count at Basel: | ine to Week 12 (BCA) | ITT Population | |
| Table 14.2.14.1 | Summary of Total Ha | ir Count at Basel | ine to Week 12 (BCA) | PP Population | |
| Table 14.2.15.1 | Summary of Total Ha | ir Count at Basel: | ine to Week 12 (WCA) | ITT Population | |
| Table 14.2.16.1 | Summary of Total Ha | ir Count at Basel: | ine to Week 12 (WCA) | PP Population | |

Table 14.2.11.2

Analysis of Change in Total Hair Count from Baseline after 12 Weeks of Treatment (LOCF)

ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| Number of patients | XXX | XXX | XXX |
| Baseline Unadjusted Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| 12 Weeks Visit | | | |
| Unadjusted Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Unadjusted Mean Change from Baseline(SE) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Adjusted Mean Change from Baseline(SE)[a] | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Versus P-3074 + P | | | |
| LS Mean Difference (SE) [a] | | x.xx (x.xxx) | |
| 95% Confidence Interval [a] | | (x.xx, x.xx) | |
| p-value [a] | | x.xxx | |

[a] The analysis uses an ANCOVA model adjusted for treatment group, center, as fixed effects and baseline hair count as a covariate. Change from Baseline by Visit is the reported result.

Program Name: Date Generated: Page x of y

| Repeat | for | the | following | displays: |
|--------|-----|-----|-----------|-----------|
|--------|-----|-----|-----------|-----------|

| Table 14.2.12.2 | Analysis of Change | in Total | Hair Count | from Baseline | after 12 V | Weeks of Treatment | (LOCF) PP Population |
|---|---|---|---|---|---|---|---|
| Table 14.2.13.2 | Analysis of Change | in Total | Hair Count | from Baseline | after 12 W | Weeks of Treatment | (BCA) ITT Population |
| Table 14.2.14.2 | Analysis of Change | in Total | Hair Count | from Baseline | after 12 W | Weeks of Treatment | (BCA) PP Population |
| Table 14.2.15.2 | Analysis of Change | in Total | Hair Count | from Baseline | after 12 W | Weeks of Treatment | (WCA) ITT Population |
| Table 14.2.16.2 | Analysis of Change | in Total | Hair Count | from Baseline | after 12 V | Weeks of Treatment | (WCA) PP Population |









Table 14.3.1.1

Overall Frequency of Patients with Adverse Events
Safety Population

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| Patients with any TEAE Patients with Mild TEAEs | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with Moderate TEAEs | xxx ( xx.x%)<br>xxx ( xx.x%) | xxx ( xx.x%)<br>xxx ( xx.x%) | xxx ( xx.x%)<br>xxx ( xx.x%) | xxx ( xx.x%)<br>xxx ( xx.x%) |
| Patients with Severe TEAEs [a] | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Study Drug Related TEAEs [a] | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any TEAE Leading to Discontinuation of Study | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Study Drug Related<br>TEAE Leading to Discontinuation of Study | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Treatment Emergent<br>Serious Adverse Events (TESAE) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Study Drug Related TESAE [b] | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any TESAE Leading to Death | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Study Drug Related<br>TESAE Leading to Death | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any TESAE Leading to Discontinuation from Study | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Patients with any Study Drug Related<br>TESAE Leading to Discontinuation from Study | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

The denominator for percentages is the number of patients in the Safety Population

Program Name: Date Generated: Page x of y

<sup>[</sup>a] Cases with unknown intensity were assumed to be severe

<sup>[</sup>b] Included are AEs considered relataed or possibly related to study drug and AEs with unknown or missing relationship to study drug

Table 14.3.1.2

Summary of Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) |
| Patients with any<br>TEAE | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| System Organ Class 1 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 1 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Preferred Term 2 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Preferred Term 3 etc. | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| System Organ Class 2 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 1 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Preferred Term 2 | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Preferred Term 3 . etc. | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) |

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Program Name: Date Generated:

Repeat for the following displays:

Generated: Page x of y

Table 14.3.1.3 Summary of Treatment-Related Treatment Emergent Adverse Events by MedDRA System Organ Class and Preferred Term Safety Population

Table 14.3.1.7 Summary of Treatment Emergent Adverse Events Causing Discontinuation from Study by MedDRA System Organ Class and Preferred Term Safety Population

Footnote: The denominator for percentages is the number of patients in the Safety Population Delete:

Footnote:

- n = number of patients in each category; The percentage is calculated as 100 x (n/N)
- e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

n = number of patients in each category; The percentage is calculated as 100 x (n/N)

e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

```
Table 14.3.1.8 Summary of Treatment-Related Treatment Emergent Adverse Events Causing Discontinuation from Study by MedDRA System Organ Class and
Preferred Term Safety Population
 Add:
   Footnote: The denominator for percentages is the number of patients in the Safety Population
  Delete:
   Footnote:
n = number of patients in each category; The percentage is calculated as 100 x (n/N)
e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)
Table 14.3.1.9 Summary of Treatment-Related Treatment Emergent Serious Adverse Events by MedDRA System Organ Class and Preferred Term Safety
Population
 Add:
   Footnote: The denominator for percentages is the number of patients in the Safety Population
  Delete:
   Footnote:
n = number of patients in each category; The percentage is calculated as 100 x (n/N)
e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)
Table 14.3.1.10
                      Summary of Adverse Events Leading to Death by MedDRA System Organ Class and Preferred Term Safety Population
  Add:
   Footnote: The denominator for percentages is the number of patients in the Safety Population
  Delete:
   Footnote:
n = number of patients in each category; The percentage is calculated as 100 x (n/N)
e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)
```

Table 14.3.1.4

Summary of Treatment Emergent Adverse Events by Relationship to Study Treatment by MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total (N = xxx) n (%)/e (%) |
|---|---|---|---|---|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) | |
| Relationship to Study Drug | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) | |
| Patients with Any TEAE | | | | |
| Overall | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Not Related | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Unlikely Related | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) |
| Possibly Related | xxx (xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Related | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| System Organ Class 1 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Not Related | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Unlikely Related | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Possibly Related | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Related | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x |
| Preferred Term 1 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Not Related | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| : | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| Preferred Term 2 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x |
| Not Related | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x |
| : | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x |
| etc | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x |

 $<sup>\</sup>mbox{\sc n}$  = number of patients in each category; The percentage is calculated as 100 x (n/N)

Program Name: Date Generated: Page x of y

e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

Note: Patients with missing relationship to study drug are counted in the Overall category only.

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term and for the episode that is most related to study drug. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Table 14.3.1.5

Summary of Treatment Emergent Adverse Events by Maximum Intensity System Organ Class and Preferred Term Safety Population

| System Organ Class | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| Maximum Severity | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) | n (%)/e (%) |
| Patients with Any | | | | |
| Maximum Intensity TEAE | | | | |
| Overall | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Mild | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Moderate | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Severe | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| System Organ Class 1 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Mild | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Moderate | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Severe | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| Preferred Term 1 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| : | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| Preferred Term 2 | | | | |
| Overall | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) |
| : | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) |
| etc | xxx(xx.x%)/xxx(xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx (xx.x%) /xxx (xx.x%) | xxx(xx.x%)/xxx(xx.x%) |

n = number of patients in each category; The percentage is calculated as 100 x (n/N)

Program Name:
Repeat for the following displays:

Date Generated:

e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

Note: Patients with missing maximum severity are considered as severe in this table.

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term and for the episode with the maximum severity. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Table 14.3.1.6 Summary of Treatment-Related Treatment Emergent Adverse Events by Maximum Intensity, System Organ Class and Preferred Term Safety Population Add:

Footnote: The denominator for percentages is the number of patients in the Safety Population
Footnote: Note: Patients with missing maximum severity are counted in the Overall category only.

Delete:
Footnote:

n = number of patients in each category; The percentage is calculated as 100 x (n/N)
e = number of episodes in each category; the percentage is calculate as 100 x (e/Total number of episodes)

Footnote: Note: Patients with missing maximum severity are considered as severe in this table.

Table 14.3.1.11
Summary of Severity Score for Skin Irritation
Safety Population

| | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) |
|---|---|---|---|
| <pre> Visit&gt;</pre> | | | |
| ermal Response | | | |
| No evidence of irritation | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| Minimal erythema, barely perceptible | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Definite erythema, readily visible; minimal oedema or minimal papular response | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Erythema and papules | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Definite oedema | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Erythema, oedema and papules | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Vescicular eruption | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Strong reaction spreading beyond test site | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Other Effects | | | |
| No other effects | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Slightly glazed appearance | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Marked glazing | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Glazing with peeling and cracking | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Glazing with fissures | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Film of dried serour exudate covering all or part of the patch site | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Small petechial erosions or scabs | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

[Repeat for all scheduled visits]

The denominator for percentages is the number of patients with non-missing data in the Safety Population for each treatment group.

Program Name: Page x of y

Table 14.3.1.12
Incidence Rate of Severity Score for Skin Irritation
Safety Population

| | | P-3074 + P $(N = xxx)$ | | Vehicle + P<br>(N = xxx) | | Vehicle + FNS<br>(N = xxx) | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Total | | | Total | | | Total | |
| | N | Time | Incidenc | N | Time | Incidence | N | Time | Incidence |
| ncidence Rate of Skin Irritation | Events | (Years) | Rate | Events | (Years) | Rate | Events | (Years) | Rate |
| Dermal Response | | | | | | | | | |
| Treatment Period | XXX | XXX | XXXX | XXX | XXX | XXXX | XXX | XXX | xxxx |
| Overall Study Period | XXX | XXX | xxxx | XXX | XXX | XXXX | XXX | XXX | XXXX |
| Other Effects | | | | | | | | | |
| Treatment Period | XXX | XXX | XXXX | XXX | XXX | XXXX | XXX | XXX | xxxx |
| Overall Study Period | XXX | XXX | XXXX | XXX | XXX | XXXX | XXX | XXX | xxxx |

Event incidence rate is calculated as the number of events interest devided by total personal time in years.

Event incidence rate is calculated as the number of events interest devided by total personal time in years. Program Name:

Date Generated:
## Table Listing 14.3.2 Serious Treatment Emergent Adverse Events Safety Population

| | | AE Line No./ | Start Date (day) | | Relationship | | Medically | SAE | |
|---|---|---|---|---|---|---|---|---|---|
| Site | Patient/<br>Age | System Organ Class/<br>Preferred Term/<br>Verbatim [a] | Stop Date (day)[b] / Duration (days) | Intensity/<br>Frequency | to Study Drug/<br>Action<br>Taken[c] | Outcome/<br>Discontinue? | Important<br>but not<br>SAE | Type<br>[d] | Comments |
| XX | xxx/xx | 1/ | DDMMMYYYY (xx) | Mild/ | Not Related/ | Resolved/ | No | 2 | |
| 2121 | mm, m | ************************************** | DDMMMYYYY (xx)<br>/xx | Single<br>Event | xxx | No | No | ٤ | |
| | | 2/<br>xxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxx | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/xx | Moderate/<br>Single<br>Event | Unlikely/<br>xxx | Death/<br>Yes | No | 3, 1 | |
| xx | xxx/xx | 1/<br>xxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxx | DDMMMYYYY (xx)/<br>Ongoing | Severe/<br>Single<br>Event | Possibly/<br>xxx | Ongoing/<br>No | No | 3 | |

- [a] Coded using MedDRA Dictionary (Version 19.0)
- [b] Relative to the day of first dose of study treatment group
- [c] Action Taken: Inc=Dose increased; No Chg=Dose not changed; Red=Dose reduced; Int=Drug interrupted; Withd=Drug withdrawn; NA=Not applicable; Un=Unknown; Oth=Other.
- [d] SAE Type: 1=Death; 2=Life Threatening; 3=Initl or Prolonged Hospitalization; 4=Persistent or Significant Disability or Incapacity; 5=Congenital Anomaly or Birth Defect.

#### Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient, start date and SOC. Program Name:

Table 14.3.4.1
Shift Table of Hematology Test Results
Safety Population

| Parameter (unit) Time point | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | $Vehicle + FNS \\ (N = xxx)$ | Overall Total (N = xxx) |
|---|---|---|---|---|
| Hematocrit (unit) | | | | |
| Week 8 | XXX | XXX | XXX | XXX |
| Baseline Low to Low | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline Low to Normal | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline Low to High | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline Normal to Low | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline Normal to Normal | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline Normal to High | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| Baseline High to Low | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline High to Normal | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Baseline High to High | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |

<Repeat for Week 24>

<Continue for Early Termination Visit>

Note: This table only presents results for patients with non-missing data at baseline and the time point of interest.

Note: Low = below lower limit of normal range, Normal = within normal limits, High = above upper limit of normal range.

Programming Notes:

Include hemoglobin, Hematology, Eosinophils, Eosinophils(%), Basophils, Basophils(%), Lymphocytes, Lymphocytes(%), Neutrophils, Neutrophils(%), Monocytes, Monocytes, Monocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration(MCHC) in the same table. Start with a new page with an analyte to be summarized.

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.3.4.2 Shift Table of Serum Chemistry Test Results Safety Population Add:

Note to Programmer: Include Alanie aminotranferase (ALT), Aspartate aminotranferase (AST), Total Bilirubin, Total Cholesterol, Triglycerides, Gamma-Glutamyltransferase (GGT), Alkaline phosphatase, Albumin, Total protein, Glucose, Creatinine, Globulin, Calcium, Potassium, Chloride, Testosterone, Sodium, Inorganic Phosphorus, Uric acid, Urea in the same table. Start with a new page with an analyte to be summarized.

Delete:

Note to Programmer: Include hemoglobin, Hematology, Eosinophils, Eosinophils(%), Basophils, Basophils(%), Lymphocytes, Lymphocytes(%), Neutrophils, Neutrophils(%), Monocytes, Monocytes(%), Erythrocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration(MCHC) in the same table. Start with a new page with an analyte to be summarized.

Table 14.3.4.3.2.1 Shift Table of Urinalysis Test Results ITT Population Note to Programmer: Include Specific Weight, pH, Leukocytes, and Erythrocytes Start with a new page with an analyte to be summarized. Delete: Note to Programmer: Include hemoglobin, Hematology, Eosinophils, Eosinophils(%), Basophils, Basophils(%), Lymphocytes, Lymphocytes(%), Neutrophils, Neutrophils (%), Monocytes, Monocytes (%), Erythrocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC) in the same table. Start with a new page with an analyte to be summarized. Footnote: Note: This table only presents results for patients with non-missing data at baseline and the time point of interest. Footnote: Note: Low = below lower limit of normal range, Normal = within normal limits, High = above upper limit of normal range. Table 14.3.4.3.2.2 Shift Table of Urinalysis Test Results Safety Population Add: Note to Programmer: Include Specific Weight, pH, Leukocytes, and Erythrocytes Start with a new page with an analyte to be summarized. Note to Programmer: Include hemoglobin, Hematology, Eosinophils, Eosinophils(%), Basophils, Basophils(%), Lymphocytes, Lymphocytes(%), Neutrophils, Neutrophils (%), Monocytes, Monocytes (%), Erythrocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC) in the same table. Start with a new page with an analyte to be summarized. Footnote: Note: This table only presents results for patients with non-missing data at baseline and the time point of interest. Footnote: Note: Low = below lower limit of normal range, Normal = within normal limits, High = above upper limit of normal range.

## Table 14.3.4.3.1.1 Shift Table of Urinalysis Test Results ITT Population

| Glucose | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| | Baseline | Baseline | Baseline | Baseline |
| | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot |
| Week 8 | | | | |
| Normal (N) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| Trace (T) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| 1+ | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| 2+ | XX XX XX XX XX XX | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | XX XX XX XX XX XX |
| 3+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 4+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| Total (Tot) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| Week 24 | | | | |
| Normal (N) | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| Trace (T) | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX XX | XX XX XX XX XX XX |
| 1+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 2+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX XX | XX XX XX XX XX XX |
| 3+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 4+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX XX | XX XX XX XX XX XX |
| Total (Tot) | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |

<Continue for Early Termination Visit>

#### Programming Notes:

Include Proteins, Glucose, Urobilinogen, and Ketones. Start with a new page with an analyte to be summarized.

For glucose, the readings are "Normal (N)", "Trace (T)", "1+", "2+", "3+", "4+".

For proteins and ketones, the readings are "Negative (-)", "Trace (T)", "1+", "2+", "3+", "4+".

For urobilinogen, the readings are "Normal (N)", "1+", "2+", "3+", "4+".

Programmers need to update the reading ranges accordingly. If there is only 5 options instead of 6 move up if display vertically and move left if displays horizontally.

Table 14.3.4.3.1.1
Shift Table of Urinalysis Test Results
ITT Population

| Protein | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| | Baseline | Baseline | Baseline | Baseline |
| | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot | N T 1+ 2+ 3+ 4+ Tot |
| Week 8 | | | | |
| Negative (-) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| Trace (T) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| 1+ | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| 2+ | xx xx xx xx xx xx xx | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 3+ | XX XX XX XX XX XX | XX XX XX XX XX XX | xx xx xx xx xx xx xx | XX XX XX XX XX XX |
| 4+ | XX XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| Total (Tot) | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx | xx xx xx xx xx xx xx |
| Week 24 | | | | |
| Negative (-) | xx xx xx xx xx xx xx | XX XX XX XX XX XX | XX XX XX XX XX XX | xx xx xx xx xx xx xx |
| Trace (T) | XX XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 1+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX XX |
| 2+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX XX | XX XX XX XX XX XX XX |
| 3+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| 4+ | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |
| Total (Tot) | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX |

<Continue for Early Termination Visit>

#### Programming Notes:

Include Proteins, Glucose, Urobilinogen, and Ketones. Start with a new page with an analyte to be summarized.

For glucose, the readings are "Normal (N)", "Trace (T)", "1+", "2+", "3+", "4+".

For proteins and ketones, the readings are "Negative (-)", "Trace (T)", "1+", "2+", "3+", "4+".

For urobilinogen, the readings are "Normal (N)", "1+", "2+", "3+", "4+".

Programmers need to update the reading ranges accordingly. If there is only 5 options instead of 6 move up if display vertically and move left if displays horizontally.

### Table 14.3.4.3.1.1 Shift Table of Urinalysis Test Results ITT Population

| Protein | P-3074 + P $(N = xxx)$ | Vehicle + P<br>(N = xxx) | Vehicle + FNS<br>(N = xxx) | Overall Total (N = xxx) |
|---|---|---|---|---|
| | Baseline | Baseline | Baseline | Baseline |
| | N 1+ 2+ 3+ 4+ Tot | N 1+ 2+ 3+ 4+ Tot | N 1+ 2+ 3+ 4+ Tot | N 1+ 2+ 3+ 4+ Tot |
| Week 8 | | | | |
| Normal (N) | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| 1+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| 2+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| 3+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| 4+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| Total (Tot) | XX XX XX XX XX | XX XX XX XX XX XX | XX XX XX XX XX XX | xx xx xx xx xx xx |
| Week 24 | | | | |
| Normal (N) | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX |
| 1+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| 2+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx |
| 3+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX |
| 4+ | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |
| Total (Tot) | xx xx xx xx xx xx | xx xx xx xx xx xx | xx xx xx xx xx xx | XX XX XX XX XX XX |

<Continue for Early Termination Visit>

Programming Notes:

Include Proteins, Glucose, Urobilinogen, and Ketones. Start with a new page with an analyte to be summarized.

For glucose, the readings are "Normal (N)", "Trace (T)", "1+", "2+", "3+", "4+".

For proteins and ketones, the readings are "Negative (-)", "Trace (T)", "1+", "2+", "3+", "4+".

For urobilinogen, the readings are "Normal (N)", "1+", "2+", "3+", "4+".

Programmers need to update the reading ranges accordingly. If there is only 5 options instead of 6 move up if display vertically and move left if displays horizontally.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

```
Table 14.3.4.3.1.2 Shift Table of Urinalysis Test Results Safety Population Delete:
```

Note to Programmer: For glucose, the readings are "Normal (N)", "Trace (T)", "1+", "2+", "3+", "4+".

For proteins and ketones, the readings are "Negative (-)", "Trace (T)", "1+", "2+", "3+", "4+".

For urobilinogen, the readings are "Normal (N)", "1+", "2+", "3+", "4+".

Programmers need to update the reading ranges accordingly. If there is only 5 options instead of 6 move up if display vertically and move left if displays horizontally.

### Table 14.3.4.3.3.1 Shift Table of Urinalysis Test Results ITT Population

| (N = xxx) $(N = xxx)$ $(N = xxx)$ $(N = xxx)$ |
|------------------------------------------------------|
| (IV AAA) (IV AAA) (IV AAA) |
| Baseline Baseline Baseline Baseline |
| Pos Neg Tot Pos Neg Tot Pos Neg Tot |
| Week 8 |
| Positive (Pos) xxx x |
| Negative (Neg) xxx x |
| Total (Tot) xxx x |
| Week 24 |
| Positive (Pos) xxx x |
| Negative (Neg) xxx x |
| Total (Tot) xxx x |

<Continue for Early Termination Visit>

Programming Notes:

Include Specific Nitrites and Bilirubin. Start with a new page with an analyte to be summarized. Program Name: Date Generated:

Repeat for the following displays:

Table 14.3.4.3.3.2 Shift Table of Urinalysis Test Results Safety Population

Table 14.3.5.1 Summary of Vital Signs ITT Population

| Weight (unit) | P-3074 + P | Vehicle + P | Vehicle + FNS |
|----------------------|---------------|---------------|----------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| Maseline | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XXX, XXX | XXX, XXX | XXX, XXX |
| Min | XX • X | XX.X | XX.X |
| Max | xx.x | XX.X | xx.x |
| <visit></visit> | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Q1, Q3 | XXX, XXX | XXX, XXX | XXX, XXX |
| Min | XX.X | XX.X | XX.X |
| Max | xx.x | XX.X | XX.X |
| Change from Baseline | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Q1, Q3 | xxx, xxx | xxx, xxx | XXX, XXX |
| Min | xx.x | xx.x | XX.X |
| Max | XX.X | XX.X | XX.X |

[Repeat for all scheduled visits]

Programming Notes:

Include Weight, Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate, and Temperature. Start with a new page with an analyte to be summarized.

Program Name:
Repeat for the following displays:

Date Generated:

Page x of y

Table 14.3.5.2 Summary of Vital Signs Safety Population

Table 14.3.6.1
Summary of Physical Exam
ITT Population

| | P-3074 + P | Vehicle + P | Vehicle + FNS | Overall Total |
|---|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) | (N = xxx) |
| creening | xxx | xxx | xxx | xxx |
| Any Abnormality?[a] | | | | |
| Normal | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal not clinically significant | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal clinically significant | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Not done | xxx ( xx.x%) | xxx ( xx.x%) | xxx (xx.x%) | xxx ( xx.x%) |
| bnormalities by Body System | | | | |
| Body System 1 | | | | |
| Normal | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal not clinically significant | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal clinically significant | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Not done | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Body System 2 | | | | |
| Normal | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal not clinically significant | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Abnormal clinically significant | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Not done | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) | xxx ( xx.x%) |
| Body System 3 | | | | |
| : | | | | |

<Repeat for all visits>

Repeat for the following displays:

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the Safety Population for each treatment group. Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in theITT Population for each treatment group.

<sup>[</sup>a] Count are based on the worst severity documented on the CRF at the visit.

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group. Program Name: Page x of y

Table 14.3.6.2 Summary of Physical Exam Safety Population

# Listing 16.2.1.1 Patients Screened All Screened Patients

Treatment group: Treatment 1

| Site | Patient/ | Date of Informed | Date of Screen | Reason(s) for Screen |
|---|---|---|---|---|
| | Age | Consent | Failure | Failure |
| XX<br>XX<br>XX | xxx/xx<br>xxx/xx<br>xxx/xx | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | Reason 1; Reason 2<br>Reason 1 |

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

Listing 16.2.1.2
Patients Disposition
All Randomized Population

| | | | Completed | Primary Reason for | Date of 1st Dose of | Date of | Date of Last Dose of |
|---|---|---|---|---|---|---|---|
| Site | Patient | Age<br>(year) | Study | Withdrawal | Study Treatment group/<br>Date of 1st Spray of<br>Study Treatment group | Withdrawal<br>(Day)[a] | Study Treatment group<br>(Day)[a]/<br>Date of Last Spray of<br>Study Treatment group |
| ΙX | XXX | xx | No | Reason 1 | DDMMMYYYY/<br>DDMMMYYYY | DDMMMYYYY (xx) | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) |
| ΚX | XXX | XX | No | Reason 2 | DDMMMYYYY/<br>DDMMMYYYY | DDMMMYYYY (xx) | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) |
| XX | XXX | XX | Yes | | DDMMMYYYY/<br>DDMMMYYYY | | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) |

[a] Relative to date of first dose of study treatment group

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient

Listing 16.2.1.3
Patients Disposition
All Randomized Population

Treatment group Group: P-3074 + P

| Site | Patient/<br>Age | Visit | Date Visit (Day)<br>[a] |
|------|-----------------|---------------|-------------------------|
| XX | xxx/xx | Screening | DDMMMYYYY (xx) |
| | | Randomization | DDMMMYYYY (xx) |
| | | Week 4 | DDMMMYYYY (xx) |
| | | Week 8 | DDMMMYYYY (xx) |
| | | Week 12 | DDMMMYYYY (xx) |

[a] Relative to date of first dose of study treatment group

Programming notes: Repeat for all treatment group groups. Sort by treatment group group, site and patient Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient

Listing 16.2.1.4
Patients Treatment Allocation
All Randomized Population

| Site | Patient/Age | Randomized<br>Treatment Group | Date of Randomization |
|------|-------------|-------------------------------|-----------------------|
| xx | xxx/xx | Treatment x | DDMMMYYYY |

Programming Notes:

Repeat for all treatment groups. Sort by site and patient Program Name: Date Generated:

Listing 16.2.1.5
Protocol Violations
All Randomized Population

Treatment group: Treatment 1

| Site | Patient/Age | Any Violations? | Date | Violation Category | Details of Violation |
|---|---|---|---|---|---|
| xx | xxx/xx | Yes<br>No | DDMMMYYYY | xxxxxxxxxxxx | xxxxxxxxxxxxxxx |

Note: Violations were identified and categorized prior to unblinding. Patients may have more than one violation leading to exclusion from All Randomized Population

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient

Listing 16.2.2.1 Inclusion Criteria All Screened Patients

Treatment group: Treatment 1

| I I Ca cin | ciic group. ircc | a CHICHE I | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site | Patient/Age | Protocol<br>Version | I1 | 12 | 13 | I4 | I5 | I6 | I7 |
| XX | xxx/xx | 1 | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| XX | xxx/xx | 1 | Yes | Yes | Yes | Yes | Yes | Yes | Yes |

Refer to Preface A for full descriptions of the Inclusion and Exclusion Criteria. Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

### Listing 16.2.2.2 Exclusion Criteria All Screened Patients

Treatment group: Treatment 1

| TTCaci | ciic group. | 11000 | IIICIIC - | L | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Patient<br>/Age | E1 | E2 | E3 | E4 | E5 | E6 | E7 | E8 | E9 | E10 | E11 | E12 | E13 | E14 | E15 | E16 | E17 | E18 |
| XX | xxx/xx | Yes | Yes | NA | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | | | | | | |
| XX | xxx/xx | No | Yes | NA | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | | | | | | |

Refer to Preface A for full descriptions of the Inclusion and Exclusion Criteria.

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

<sup>[</sup>a] Relative to the day of first dose of study treatment group

Listing 16.2.3 Study Population All Screened Patients

Treatment group: Treatment 1 Patient/ All Screened All Safety ITT Per Protocol Age Patient Randomized Population Population Population Population xxx/xx Yes XX Yes Yes Yes Yes xxx/xxYes Yes Yes No No XX

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

# Listing 16.2.4.1 Demographics All Randomized Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Year of Birth | Race | Ethnicity | Current Tobacco<br>Use/<br>Smoke>=10<br>cigerretts per day | Current Alocohol<br>Use | Drink>5 Cups of coffee/tea per day |
|---|---|---|---|---|---|---|---|
| xx | xxx/xx | YYYY | Race1 | Ethnicity1 | Never/No | None | Yes |
| XX | xxx/xx | YYYY | Race2 | Ethnicity2 | Current/No | <=2 drinks per day | Yes |
| XX | xxx/xx | YYYY | Other: xxxx | Ethnicity3 | Former/Yes | > 2 drinks per day | No |

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

Listing 16.2.4.2 Medical History All Randomized Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Vertex Pattern | System Organ Code (SOC)/<br>Preferred Term (PT)[a]/<br>Verbatim/<br>MMH Line No. | Start Date/<br>Stop Date[b] |
|---|---|---|---|---|
| XX | xxx/xx | Type III | xxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxx/<br>xxxxxx | DDMMMYYYY/<br>DDMMMYYYY |
| XX | xxx/x | Type IV | xxxxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxxx | DDMMMYYY/<br>Ongoing |
| XX | xxx/xx | Other: xxxxx | None | |

[a] MedDRA Dictionary (Version 19.0) was used for coding Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient, SOC and preferred term. Program Name:

Date Generated:

## Listing 16.2.4.3 Prior and Concomitant Medication All Randomized Population

Treatment group: Treatment 1

| Site | Patient<br>/Age | Therapeutic Class<br>Chemical Subgroup<br>Generic Term [a] | Dose/Unit/<br>Frequency/<br>Route | Indication<br>CM Number | Start Date (day) Stop Date (day)[b] / Duration (days) |
|---|---|---|---|---|---|
| xx | xxx/xx | xxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxx | xx/units/<br>xx/<br>xx | xxxxxxxxx<br>xx, xx /1 | DDMMMYYYY (xx)<br>DDMMMYYYY (xx)<br>/xx |
| | | xxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxx | xx/units/<br>xx/<br>xx | xxxxxxxxx<br>xx, xx /2 | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/xx |
| xx | xxx/xx | xxxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxx | xx/units/<br>xx/<br>xx | xxxxxxxxx<br>xx, xx /1 | DDMMMYYYY (xx)/<br>Ongoing |
| XX | xxx/xx | None | | | |

Repeat for all treatment groups. Sort by treatment group, site, patient, start date and drug class. Program Name:

Date Generated:

<sup>[</sup>a] WHO Drug Dictionary (Version MAR16B2E) was used for coding

<sup>[</sup>b] Relative to date of first dose of study treatment group

Programming Notes:

# Listing 16.2.5.1 Study Drug Administration (Tablet) All Randomized Population

Treatment group Group: P-3074 + P

| Site | Patient/<br>Age | Start Date<br>Time of<br>Treatment | Last Date Time<br>of Treatment | Start Date of<br>Interruption<br>(day) [a] | End Date of Interruption (day) [a] | Actual<br>Treatment<br>Received |
|---|---|---|---|---|---|---|
| xx | xxx/xx | DDMMMYYYY<br>HH:MM | DDMMMYYYY HH:MM | DDMMMYYYY (xx) | DDMMMYYYY (xx) | xxxxx |

[a] Relative to the day of first dose of study treatment group Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

### Listing 16.2.5.2 Study Drug Administration (Spray) All Randomized Population

Treatment group Group: P-3074 + P

| Site | Patient/<br>Age | Start Date<br>Time of<br>Treatment | Last Date Time<br>of Treatment | Start Date of<br>Interruption<br>(day) [a] | End Date of<br>Interruption (day)<br>[a] | Actual<br>Treatment<br>Received |
|---|---|---|---|---|---|---|
| xx | xxx/xx | DDMMMYYYY<br>HH:MM | DDMMMYYYY HH:MM | DDMMMYYYY (xx) | DDMMMYYYY (xx) | xxxxxx |

[a] Relative to the day of first dose of study treatment group Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient Program Name:

Date Generated:

# Listing 16.2.5.3 Study Treatment Compliance/Exposure All Randomized Population

Treatment group: Treatment 1

| | | Compliance | Based on Diary | Compliance Ba | sed Accountability | |
|---|---|---|---|---|---|---|
| Site | Patient/ | Tablets (%) | Spray Shot (%) | Tablets (%) | Spray Shot (%) | Duration of |
| | Age | | | | | Exposure (days) |
| XX | xxx/xx | XX.X% | XX.X% | XX.X% | XX.X% | XXXX |

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient and visit. Program Name:

Date Generated:

Listing 16.2.6.1 Hair Assessment Results All Randomized Population

Treatment group: Treatment 1

| I I Ca cin | cne group. rrea | CINCII C | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Site | Patient/Age | Visit | Date (day)<br>[a] | Hair Count | Hair Wi<br>(unit) | ldth | | | | | |
| XX | xxx/xx | | | 10 | 10.36<br>7.55 | 12.23<br>8.65 | 13.15<br>8.99 | 8.33 | 6.45 | 9.32 | 6.88 |

[a] Relative to the day of first dose of study treatment group

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site and patient

Please include all measured hair width in this listing.

### Listing 16.2.6.2 MHGQ Questionnaire All Randomized Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Visit | Collection<br>Data(day) [a] | Question | Patient's Response/Score |
|---|---|---|---|---|---|
| xx | xxx/xx | Week 12 | DDMMMYYYY (xx) | Bald spot getting smaller? Appreance of my hair is: Growth of my hair Effctive of the treatment Hairline at the frond Hair on top Overall | Agree/2 A littie better/3 Slightly increased/3 Somehow effective/2 I am very satisfied/1 I am satisfied/2 I am satisfied/2 |

[a] Relative to the day of first dose of study treatment group

Listing 16.2.6.3

Blind Assessor Assessment of Patient Hair Growth/Loss Change from Baseline
All Randomized Population

Treatment group: Treatment 1

| TTCacin | ciic group. | II Ca chiche I | | |
|---|---|---|---|---|
| Site | Patient/<br>Age | Visit | Assessment<br>Data(day) [a] | Assessment of Hair Growth |
| XX | xxx/xx | Week 12<br>Week 24 | DDMMMYYYY (xx)<br>DDMMMYYYY (xx) | Greatly Increased Greatly Increased |

[a] Relative to the day of first dose of study treatment group

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Listing 16.2.6.4 Investigator's Assessment of Patient Hair Growth/Loss Change from Baseline All Randomized Population

Delete:

Footnote: [a] Relative to the day of first dose of study treatment group



Listing 16.2.7.1 Adverse Events Safety Population

| Treatm | ent group: | Treatment 1 | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site | Patient/<br>Age | AE Line No./<br>System Organ Class/<br>Preferred Term/<br>Verbatim [a] | TEAE or PTAE/<br>Start Date (day)<br>Stop Date (day)[b]<br>/ Duration (days) | Intensity/<br>Frequency | Relationship<br>to Study Drug/<br>Action<br>Taken[c] | Outcome/<br>Discontinue? | Medically<br>Important<br>but not<br>SAE | SAE[d] | Comments |
| xx | xxx/xx | 1/<br>xxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxx | TEAE/ DDMMMYYYY (xx) DDMMMYYYYY (xx) /xx | Mild/<br>Single<br>Event | Not Related/<br>xxx | Resolved/<br>No | No | No | |
| | | 2/<br>xxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxx/<br>xxxxxx | TEAE/ DDMMMYYYY (xx)/ DDMMMYYYY (xx)/xx | Moderate/<br>Single<br>Event | Unlikely/<br>xxx | Death/<br>Yes | No | Yes:1 | |

[a] Coded using MedDRA Dictionary (Version 19.0)

xxxxxxxxxxxxxxxx/

xxxxxxxxxxxxxx/

[b] Relative to the day of first dose of study treatment group

PTAE/

Ongoing

[c] Action Taken: Inc=Dose increased; No Chg=Dose not changed; Red=Dose reduced; Int=Drug interrupted; Withd=Drug withdrawn; NA=Not applicable; Un=Unknown; Oth=Other

Severe/

Single

Event

Not Related/

XXX

Ongoing/

[d] SAE Type: 1=Death; 2=Life Threatening; 3=Initl or Prolonged Hospitalization; 4=Persistent or Significant Disability or Incapacity; 5=Congenital Anomaly or Birth Defect

Programming Notes:

XX

xxx/xx 1/

Repeat for all treatment groups. Sort by treatment group, site, patient, start date and SOC.

Program Name:

Date Generated:

Page x of y

Yes:3

Repeat for the following displays:

Listing 16.2.7.2 Treatment Emergent Adverse Events Leading to Discontinuation of Treatment Safety Population

Listing 16.2.7.3 Death Safety Population

# Listing 16.2.7.4 Severity Score for Skin Irritation Safety Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Visit | Collection<br>Data(day) [a] | Dermal Response | Other Effects |
|---|---|---|---|---|---|
| xx | xxx/xx | Week 4<br>Week 8<br>Week 12<br>Week 24<br>Week 28 | DDMMMYYYY (xx) DDMMMYYYY (xx) DDMMMYYYY (xx) DDMMMYYYY (xx) | No evidence of irritation Erythema and papules Erythema, oedema and papules Vescicular eruption Strong reaction spreading beyond test site | No other effetcs Marked glazing Marked glazing Slight glazed appearance No other effetcs |
| XX | xxx/xx | Week 4 | DDMMMYYYY (xx) : : | No evidence of irritation: : : | No other effetcs : : : |

Listing 16.2.8.1
Preface to Laboratory Findings
Safety Population

| Laboratory Test | Sex | Age | Reference Ranges | Unit |
|-----------------|-----|-----|-------------------|--------|
| Hematology | | | xxxxxxx - xxxxxxx | |
| Hematocrit | | | | (unit) |
| Hemoglobin | | | | (unit) |
| Serum Chemistry | | | | |
| ALT | | | | (unit) |
| AST | | | | (unit) |

#### Listing 16.2.8.2 Laboratory Findings - Hematology Safety Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Nominal<br>Visit | Laboratory<br>Parameter<br>(unit) | Collection Date (day) [a] | Was Blood<br>Sample<br>Collected? | Value [b] | Normal<br>Range | Overall<br>Evaluation |
|---|---|---|---|---|---|---|---|---|
| XX | xxx/xx | Screening | Hematocrit | DDMMMYYYY (xx) | Yes | xxx.xxx B | xxx - xxx | Normal |
| | | Week 8 | Hematocrit | DDMMMYYYY (xx) | Yes | XXX.XXX | xxx - xxx | Normal |
| | | Week 24 | Hematocrit | DDMMMYYYY (xx) | Yes | XXX.XXX | xxx - xxx | Abnormal not clinically significant |
| | | ETV | : | : | : | : | : | : |
| | | : | : | : | : | : | : | : |
| | | Screening | Hemoglobin | DDMMMYYYY (xx) | Yes | xxx.xxx A | xxx - xxx | : |
| | | Week 8 | Hemoglobin | DDMMMYYYY (xx) | Yes | XXX.XXX | xxx - xxx | : |
| | | Week 24 | Hemoglobin | DDMMMYYYY (xx) | Yes | XXX.XXX | xxx - xxx | Abnormal not clinically significant |
| | | : | : | : | : | : | : | : |
| | | : | : | : | : | : | : | |
| | | | Continue for | all Hematology pa | rameters | | | |

<sup>[</sup>a] Relative to the day of first dose of study treatment group

Programming Notes:

Include Hematocrit, Hemoglobin, White Blood Cell Count with Differential (Eosinophils,

Basophils, Lymphocytes, Neutrophils, Monocytes), Erythrocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean

Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC)

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Listing 16.2.8.3 Laboratory Findings - Serum Chemistry Safety Population

Add:

Note to Programmer: Include Alanine aminotranferase (ALT), Aspartate aminotranferase (AST), Total Bilirubin, Total Cholesterol, Triglycerides, Gamma-Glutamyltransferase (GGT), Alkaline phosphatase, Albumin, Total protein

Glucose, Creatinine, Globulin, Calcium, Potassium, Chloride, Testosterone, Sodium, Inorganic Phosphorus, Uric acid, Urea Delete:

Note to Programmer: Include Hematocrit, Hemoglobin, White Blood Cell Count with Differential (Eosinophils,

Basophils, Lymphocytes, Neutrophils, Monocytes), Erythrocytes, Thrombocytes, Mean Corpuscular Volume (MCV), Mean Corpuscular hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC)

<sup>[</sup>b] B=Below, A=Above the normal limits

## Listing 16.2.8.4 Laboratory Findings - Urinalysis Safety Population

Treatment group: Treatment 1

| Site | Patient/Age | Nominal<br>Visit | Laboratory<br>Parameter<br>(unit) | Collection<br>Date (day) | [a] | Was Urine<br>Sample<br>Collected? | Value | Overall<br>Inspection |
|---|---|---|---|---|---|---|---|---|
| xx | xxx/xx | Screening<br>Week 8 | PH<br>PH | • | xx) | Yes<br>Yes | XXX | Normal<br>Normal |
| | | Week 24 | PH | , | xx) | Yes | XXX | Abnormal not clinically significant |
| | | ETV | : | : | | : | : | : |
| | | : | : | : | | : | : | : |
| | | Screening | Color | DDMMMYYYY (: | xx) | Yes | XXX | : |
| | | Week 8 | Color | DDMMMYYYY (: | xx) | Yes | XXX | : |
| | | Week 24 | Color | DDMMMYYYY (: | xx) | Yes | XXX | Abnormal not clinically significant |
| | | : | : | : | | : | : | : |
| | | : | : | : | | : | : | |
| | | | Continue for | all Urinalysi | is pa | rameters | | |

[a] Relative to the day of first dose of study treatment group Programming Notes:

Include Macroscopic analysis: pH, specific weight, appearance, colour, nitrites, proteins, glucose, urobilinogen, bilirubin, ketones, haematic pigments, leukocytes
Microscopic analysis: leukocytes, Erythrocytes, flat cells, round cells, crystals, cylinders, mucus, bacteria

Listing 16.2.8.5 Vital Signs Safety Population

Treatment group: Treatment 1

| Site | Patient/<br>Age | Nominal<br>Visit | Collection<br>Date (day) [a] | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m²) | SBP<br>(mmHg) | DBP<br>(mmHg) | Pulse<br>(bpm) | Temperature (C) |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | xxx/xx | Screening<br>Week 24<br>Week 28 | DDMMMYYYY(xx)<br>DDMMMYYYY(xx)<br>DDMMMYYYY(xx) | xxxxx<br>xxxxx<br>xxxxx | xxxxx<br>xxxxx<br>xxxxx | xxxx<br>xxxx<br>xxxx | xxxx<br>xxxx<br>xxxx | XXXX<br>XXXX | xxxx<br>xxxx<br>xxxx | xxx<br>xxx<br>xxx |

Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient and visit. Temperature is collected in 2 units. Please convert F to C.  $T(^{\circ}C) = (T(^{\circ}F) - 32) \times 5/9$ Program Name:

Date Generated: Page x of y

<sup>[</sup>a] Relative to the day of first dose of study treatment group

Note: Body temperature is reported in Celsius. For those patients who reported their body temperature in Fahrenheit. The following coversion will be used:  $T(^{\circ}C) = (T(^{\circ}F) - 32) \times 5/9$ 

Listing 16.2.8.6
Physical Examination Results
Safety Population

Treatment group: Treatment 1

| | Patient/ | | Assessment Date (day) | Body System | |
|---|---|---|---|---|---|
| Site | Age | Visit | [a] | Abnormalities | Findings |
| XX | xxx/xx | Baseline | DDMMMYYYY (xx) | Cardiovascular | xxxxxxxxxxxxxxx |
| | | | , , | Respiratory | XXXXXXXXXXXXXXXX |
| | | | | Gastrointestinal | XXXXXXXXXXXXXXXX |
| | | | | Skin | XXXXXXXXXXXXXXXX |
| | | | | Musculoskeletal | XXXXXXXXXXXXXXX |
| | | | | Endocrine | XXXXXXXXXXXXXXXX |
| | | | | Neurological | XXXXXXXXXXXXXXX |
| | | | | HEENT | XXXXXXXXXXXXXXX |
| | | | | Genitourinary | XXXXXXXXXXXXXXX |
| | | Week x | DDMMMYYYY (xx) | None | Patient refusal |

[a] Relative to the day of first dose of study treatment group Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient and visit. Only present abnormal body systems. If all body systems are normal at a visit, output "None" in Body System Abnormalities column for the visit.

If PE is not performed, please display "No PE performed" under Body System Abnormalities column and report reason not performed under "Findings" column.

### Listing 16.2.8.7 Self-administered Sexual Dysfunction Questionnaire Safety Population

Treatment group: Treatment 1

| | Patient/ | | Assessment Date (day) | | |
|---|---|---|---|---|---|
| Site | Age | Visit | [a] | Question: Over the past 4 weeks | Answer |
| xx x | xxx/xx | Week 4 | DDMMMYYYY (xx) | How often were you able to get an erection during sexual activity? | No sexual activity |
| | | | | When you had erections with sexual stimulation, how often were your erections hard enough for penetration? | Almost always or always |
| | | | | When you attempted sexual intercourse how often were you able to penetrate (enter) your partner? | Most times |
| | | | | During sexual intercourse how often were you able to maintain your erection after you had penetrated (entered) your partner? | Did not attempt intercourse |
| | | | | During sexual intercourse how difficult was it to maintain your erection to completion of intercourse? | Slightly difficul |
| | | | | :<br>: | : |
| | | Week 8 | DDMMMYYYY (xx) | How often were you able to get an erection during sexual activity? | No sexual activit |
| | | | | : | : |
| | | | | : | : |

[a] Relative to the day of first dose of study treatment group Programming Notes:

Repeat for all treatment groups. Sort by treatment group, site, patient and visit.

Figure 14.1.6
Study Treatment Compliance
ITT Population



 $\mbox{Figure 14.2.1.1} \\ \mbox{Hair Count Unadjusted Mean Change From Baseline by Treatment Over Time } \\ \mbox{ITT Population}$ 



Note: Vertical bar represents 95% CI.

Program Name:

Repeat for the following displays:
Figure 14.2.1.2 Hair Count Adjusted Mean Change From Baseline by Treatment Over Time ITT Population

Figure 14.2.2.1 Hair Count Unadjusted Mean Change From Baseline by Treatment Over Time PP Population

Figure 14.2.2.2 Hair Count Adjusted Mean Change From Baseline by Treatment Over Time PP Population

Figure 14.2.3.1 Hair Width Unadjusted Mean Change From Baseline by Treatment Over Time ITT Population

Figure 14.2.3.2 Hair Width Adjusted Mean Change From Baseline by Treatment Over Time ITT Population

| Figure 14.2.4.1 | Hair Width | Unadjusted Mea | n Change Fr | om Baseline b | y Treatment | Over Time PA | Population |
|---|---|---|---|---|---|---|---|
| Figure 14.2.4.2 | Hair Width | Adjusted Mean | Change From | Baseline by | Treatment Ov | ver Time PP I | Population |

Figure 14.2.8.1
Unadjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time ITT Population



Program Name:

Repeat for the following displays:
Figure 14.2.8.2 Adjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time

Figure 14.2.9.1 Unadjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time

Propulation

Figure 14.2.9.2 Adjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time

Propulation

Adjusted Investigator Assessment of Improvement Patient Hair Growth/Loss Mean Score from Baseline by Treatment Over Time

Propulation

